CLINICAL TRIAL: NCT00423046
Title: Phase IIIb, Observer-blind Study to Compare Immunogenicity of GSK Biologicals' HPV-16/18 L1/AS04 Vaccine Versus Gardasil® [Quadrivalent Human Papillomavirus (HPV-6,11,16,18 L1 VLP) Recombinant Vaccine Merck & Co., Inc.]
Brief Title: Immunogenicity of GlaxoSmithKline Biological's Human Papillomavirus (HPV) Vaccine (580299) Versus Merck's Gardasil® in Healthy Females 18-45 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 108933
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Results first posted 2010-08-25 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Infections, Papillomavirus; Papillomavirus Vaccines
Keywords: Vaccines; Cervical cancer; Immunogenicity; Humans; Safety; Viral infections; Human papillomavirus (HPV); Comparative study; Human papillomavirus vaccine; Adults
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Virus Diseases | interventions — human papillomavirus vaccine, L1 type 16, 18; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Cervarix Group (Experimental): Subjects received 3 doses of GSK Biologicals human papillomavirus [HPV]16/18 vaccine 580299 (CervarixTM) at Months 0, 1 and 6 and a dose of placebo at Month 2. All doses were administered by intramuscular injection in the deltoid muscle of the upper arm.
  Interventions: Biological: GSK Biologicals HPV 16/18 vaccine 580299 (CervarixTM); Biological: Placebo
- Gardasil Group (Active Comparator): Subjects received 3 doses of Gardasil® (Merck's human papillomavirus [HPV] vaccine) at Months 0, 2 and 6 and a dose of placebo at Month 1. All doses were administered by intramuscular injection in the deltoid muscle of the upper arm.
  Interventions: Biological: Gardasil ® (Merck & Co. Inc); Biological: Placebo

INTERVENTIONS:
Biological: GSK Biologicals HPV 16/18 vaccine 580299 (CervarixTM) — Three doses administered intramuscularly at months 0, 1 and 6
  Other Names: Cervarix
  Arms: Cervarix Group
Biological: Gardasil ® (Merck & Co. Inc) — Three doses administered intramuscularly at months 0, 2 and 6
  Arms: Gardasil Group
Biological: Placebo — One dose administered intramuscularly at month 1 to maintain blinding
  Arms: Gardasil Group
Biological: Placebo — One dose administered intramuscularly at month 2 to maintain blinding
  Arms: Cervarix Group

SUMMARY:
HPV infection has been established as a necessary cause of cervical cancer. GSK Biologicals has developed an HPV-16/18 L1 VLP AS04 vaccine (Cervarix TM) which targets the 2 most common oncogenic HPV types (HPV-16 and HPV-18), found in > 70%, approximately, of all cervical cancers. Recently, Merck's HPV vaccine Gardasil® [quadrivalent human papillomavirus (HPV-6,11,16,18 L1 VLP) recombinant vaccine] has been approved by the FDA for prevention of genital tract cancers and pre-cancers and genital warts in females. Although the GSK HPV vaccine and Gardasil® have different compositions and are expected to have different efficacy profiles, each vaccine targets prevention of HPV-16 and 18 genital tract cancers and pre-cancers. Therefore, a comparison of the immunogenicity of the two vaccines is warranted. This Phase 3b study is designed to compare the immunogenicity of the GSK vaccine (HPV-16/18) to Gardasil® in healthy adult females 18-45 years of age.

The Protocol Posting has been updated as the study will be extended by 3 additional years.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol Amendment 25, November 2010

ELIGIBILITY:
Inclusion Criteria:

* A woman whom the investigator believes that she or her legally acceptable representative (in the event that the subject is illiterate) can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits).
* A woman between and including 18 and 45 years of age at the time of the first vaccination.
* Written informed consent must be obtained from the subject prior to enrollment.
* Subject must be free of obvious health problems as established by medical history and history-directed clinical examination before entering into the study.
* Subject must have a negative urine pregnancy test.
* Subject must be of non-childbearing potential, or if she is of child bearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.
* Subject must have an intact cervix.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period up to Month 60.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose or planned administration during the study period up to Month 60.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after (i.e. days 0-29) each dose of vaccine. Administration of routine vaccines up to 8 days before each dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Pregnant or breastfeeding. Women must be at least 3 months post-pregnancy and not breastfeeding to enter the study.
* A woman planning to become pregnant or planning to discontinue contraceptive precautions during approximately the first eight months of the study (Months 0-8).
* Previous administration of components of the investigational vaccine
* Previous or planned vaccination against HPV outside of this protocol.
* Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccines.
* Hypersensitivity to latex.
* Known acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* History of significant medical conditions and currently under treatment.
* Received immunoglobulins and/or blood product within 90 days preceding enrolment or planned administration during the study period up to Month 60. Enrollment will be deferred until the subject is outside of specified window.
* Acute disease at the time of enrolment. Enrollment will be deferred until condition is resolved. All vaccines can be administered to persons with a minor illness
* Heavy bleeding (menstruation or other) or heavy vaginal discharge in which a pelvic exam cannot be performed. Enrollment will be deferred until condition is resolved according to investigator's medical judgement.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1106 (Actual)
Dates: Start 2007-01-24 (Actual); Primary Completion 2008-03-07 (Actual); Study Completion 2012-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (39):
- United States (39):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Louisville, Colorado
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Willoughby Hills, Ohio
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Upper Saint Clair, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Walla Walla, Washington
  - GSK Investigational Site, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=206

REFERENCES:
- [Background] Coursaget P et al. (2011) Priming as a basis for long-term protection and implications for HPV vaccination. Gynecologic Oncology. 121:S1-S9.
- [Background] Einstein MH, Baron M, Levin MJ, Chatterjee A, Edwards RP, Zepp F, Carletti I, Dessy FJ, Trofa AF, Schuind A, Dubin G; HPV-010 Study Group. Comparison of the immunogenicity and safety of Cervarix and Gardasil human papillomavirus (HPV) cervical cancer vaccines in healthy women aged 18-45 years. Hum Vaccin. 2009 Oct;5(10):705-19. doi: 10.4161/hv.5.10.9518. Epub 2009 Oct 14. PMID 19684472
- [Background] Einstein MH, Baron M, Levin MJ, Chatterjee A, Fox B, Scholar S, Rosen J, Chakhtoura N, Meric D, Dessy FJ, Datta SK, Descamps D, Dubin G; HPV-010 Study Group. Comparative immunogenicity and safety of human papillomavirus (HPV)-16/18 vaccine and HPV-6/11/16/18 vaccine: follow-up from months 12-24 in a Phase III randomized study of healthy women aged 18-45 years. Hum Vaccin. 2011 Dec;7(12):1343-58. doi: 10.4161/hv.7.12.18281. Epub 2011 Dec 1. PMID 22048173
- [Background] Einstein MH, Baron M, Levin MJ, Chatterjee A, Fox B, Scholar S, Rosen J, Chakhtoura N, Lebacq M, van der Most R, Moris P, Giannini SL, Schuind A, Datta SK, Descamps D; HPV-010 Study Group. Comparison of the immunogenicity of the human papillomavirus (HPV)-16/18 vaccine and the HPV-6/11/16/18 vaccine for oncogenic non-vaccine types HPV-31 and HPV-45 in healthy women aged 18-45 years. Hum Vaccin. 2011 Dec;7(12):1359-73. doi: 10.4161/hv.7.12.18282. Epub 2011 Dec 1. PMID 22048172
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Background] Coursaget P et al. (2011) Priming as a basis for long-term protection and implications for HPV vaccination. Gynecologic Oncology . 121:S1-S9.
- [Background] Einstein MH, Levin MJ, Chatterjee A, Chakhtoura N, Takacs P, Catteau G, Dessy FJ, Moris P, Lin L, Struyf F, Dubin G; HPV-010 Study Group. Comparative humoral and cellular immunogenicity and safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine and HPV-6/11/16/18 vaccine in healthy women aged 18-45 years: follow-up through Month 48 in a Phase III randomized study. Hum Vaccin Immunother. 2014;10(12):3455-65. doi: 10.4161/hv.36117. PMID 25483700
- [Background] Einstein MH, Takacs P, Chatterjee A, Sperling RS, Chakhtoura N, Blatter MM, Lalezari J, David MP, Lin L, Struyf F, Dubin G; HPV-010 Study Group. Comparison of long-term immunogenicity and safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine and HPV-6/11/16/18 vaccine in healthy women aged 18-45 years: end-of-study analysis of a Phase III randomized trial. Hum Vaccin Immunother. 2014;10(12):3435-45. doi: 10.4161/hv.36121. PMID 25483701
- [Background] Schwarz TF, Kocken M, Petaja T, Einstein MH, Spaczynski M, Louwers JA, Pedersen C, Levin M, Zahaf T, Poncelet S, Hardt K, Descamps D, Dubin G. Correlation between levels of human papillomavirus (HPV)-16 and 18 antibodies in serum and cervicovaginal secretions in girls and women vaccinated with the HPV-16/18 AS04-adjuvanted vaccine. Hum Vaccin. 2010 Dec;6(12):1054-61. doi: 10.4161/hv.6.12.13399. Epub 2010 Dec 1. PMID 21157180
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 108933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108933 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who missed Month 7 visit and/or one or more follow-up visits were permitted to attend the next scheduled follow-up visits.
Groups:
- Cervarix Group: Subjects received 3 doses of GSK Biologicals human papillomavirus [HPV] 16/18 vaccine 580299 (CervarixTM) at Months 0, 1 and 6 and a dose of placebo at Month 2. All doses were administered by intramuscular injection in the deltoid muscle of the upper arm.
Period: Overall Study
Arm/Group | Cervarix Group | Gardasil Group
Started | 553 | 553
Completed | 213 (Completed until Month 60) | 208 (Completed until Month 60)
Not Completed | 340 | 345
Not completed — Other | 340 | 345

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Gardasil Group | Total
Number analyzed (Participants) | 553 | 553 | 1106
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (8.02) | 30.2 (7.78) | 30.25 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 553 | 553 | 1106
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Neutralizing Antibodies
Description: Titers are displayed as Geometric Mean Titers (GMTs). The titer is the serum dilution giving a 50 percent reduction of the signal compared to a control without serum.
Time Frame: At Month 7
Population: Analysis was performed on subjects from the According-to-Protocol (ATP) cohort for immunogenicity aged 18 to 26 years and who were seronegative by Pseudovirion (PSV) neutralizing assay and deoxyribonucleic acid (DNA) negative for the corresponding type at baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 118 | 131
titer
  Anti-HPV-16: number analyzed (Participants) | 104 | 103
  Anti-HPV-16 | 36791.8 [29265.6 to 46253.6] | 10053.1 [8135.8 to 12422.1]
  Anti-HPV-18 | 16486.9 [13383.4 to 20310.1] | 2257.9 [1809.4 to 2817.7]

2. Secondary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Neutralizing Antibodies
Description: Titers are given as Geometric Mean Titers (GMTs). Titer is the serum dilution giving a 50 percent reduction of the signal compared to a control without serum.
  Data for Month 7 on subjects aged 18 to 26 years are given in the outcome above as a primary outcome measure.
Time Frame: At Month 6, 7, 12, 18, 24, 36, 48 and 60
Population: Analysis was performed by age group on subjects from the According-to-Protocol (ATP) cohort for immunogenicity who were seronegative by Pseudovirion neutralizing assay and deoxyribonucleic acid (DNA) negative for the corresponding type at baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 118 | 130
Titer
  Anti-HPV-16, 18-26-year, Month 6: number analyzed (Participants) | 104 | 102
  Anti-HPV-16, 18-26-year, Month 6 | 1627.9 [1304.0 to 2032.3] | 1592.4 [1204.3 to 2105.7]
  Anti-HPV-16, 18-26-year, Month 12: number analyzed (Participants) | 101 | 99
  Anti-HPV-16, 18-26-year, Month 12 | 14524.7 [11069.7 to 19058.0] | 3265.2 [2544.7 to 4189.7]
  Anti-HPV-16, 18-26-year, Month 18: number analyzed (Participants) | 100 | 91
  Anti-HPV-16, 18-26-year, Month 18 | 6000.3 [4681.2 to 7691.0] | 1182.7 [882.7 to 1584.8]
  Anti-HPV-16, 18-26-year, Month 24: number analyzed (Participants) | 97 | 89
  Anti-HPV-16, 18-26-year, Month 24 | 5184.2 [4015.0 to 6693.8] | 893.5 [672.2 to 1187.9]
  Anti-HPV-16, 18-26-year, Month 36: number analyzed (Participants) | 60 | 62
  Anti-HPV-16, 18-26-year, Month 36 | 3844.7 [2803.6 to 5272.3] | 653.2 [460.4 to 926.7]
  Anti-HPV-16, 18-26-year, Month 48: number analyzed (Participants) | 54 | 57
  Anti-HPV-16, 18-26-year, Month 48 | 3900.9 [2745.4 to 5542.6] | 750.4 [505.1 to 1114.8]
  Anti-HPV-16, 18-26-year, Month 60: number analyzed (Participants) | 35 | 40
  Anti-HPV-16, 18-26-year, Month 60 | 4117.8 [2742.1 to 6183.7] | 529.8 [343.2 to 817.9]
  Anti-HPV-16, 27-35-year, Month 6: number analyzed (Participants) | 90 | 84
  Anti-HPV-16, 27-35-year, Month 6 | 1263.1 [892.7 to 1787.2] | 1014.1 [737.6 to 1394.1]
  Anti-HPV-16, 27-35-year, Month 7: number analyzed (Participants) | 90 | 85
  Anti-HPV-16, 27-35-year, Month 7 | 23907.9 [18912.7 to 30222.4] | 4958.4 [3895.6 to 6311.2]
  Anti-HPV-16, 27-35-year, Month 12: number analyzed (Participants) | 91 | 85
  Anti-HPV-16, 27-35-year, Month 12 | 7419.2 [5592.1 to 9843.3] | 1755.9 [1290.3 to 2389.7]
  Anti-HPV-16, 27-35-year, Month 18: number analyzed (Participants) | 87 | 83
  Anti-HPV-16, 27-35-year, Month 18 | 2907.9 [2229.2 to 3793.1] | 689.8 [505.8 to 940.8]
  Anti-HPV-16, 27-35-year, Month 24: number analyzed (Participants) | 84 | 79
  Anti-HPV-16, 27-35-year, Month 24 | 2269.2 [1765.8 to 2916.2] | 618.8 [447.4 to 856.0]
  Anti-HPV-16, 27-35-year, Month 36: number analyzed (Participants) | 63 | 49
  Anti-HPV-16, 27-35-year, Month 36 | 1897.6 [1418.9 to 2537.8] | 501.7 [346.7 to 726.0]
  Anti-HPV-16, 27-35-year, Month 48: number analyzed (Participants) | 54 | 51
  Anti-HPV-16, 27-35-year, Month 48 | 2046.3 [1469.4 to 2849.8] | 677.6 [433.0 to 1060.2]
  Anti-HPV-16, 27-35-year, Month 60: number analyzed (Participants) | 43 | 29
  Anti-HPV-16, 27-35-year, Month 60 | 1925.3 [1301.9 to 2847.4] | 346.4 [214.9 to 558.4]
  Anti-HPV-16, 36-45-year, Month 6: number analyzed (Participants) | 96 | 81
  Anti-HPV-16, 36-45-year, Month 6 | 1729.8 [1214.8 to 2463.1] | 1916.5 [1361.3 to 2698.2]
  Anti-HPV-16, 36-45-year, Month 7: number analyzed (Participants) | 96 | 83
  Anti-HPV-16, 36-45-year, Month 7 | 17301.5 [13605.3 to 22001.9] | 7634.4 [5915.7 to 9852.5]
  Anti-HPV-16, 36-45-year, Month 12: number analyzed (Participants) | 89 | 83
  Anti-HPV-16, 36-45-year, Month 12 | 7110.4 [5386.3 to 9386.4] | 2678.2 [1986.8 to 3610.2]
  Anti-HPV-16, 36-45-year, Month 18: number analyzed (Participants) | 90 | 82
  Anti-HPV-16, 36-45-year, Month 18 | 2344.0 [1807.7 to 3039.4] | 994.8 [732.9 to 1350.4]
  Anti-HPV-16, 36-45-year, Month 24: number analyzed (Participants) | 87 | 80
  Anti-HPV-16, 36-45-year, Month 24 | 2058.5 [1592.2 to 2661.3] | 874.7 [636.9 to 1201.3]
  Anti-HPV-16, 36-45-year, Month 36: number analyzed (Participants) | 61 | 57
  Anti-HPV-16, 36-45-year, Month 36 | 1794.2 [1278.1 to 2518.8] | 823.7 [567.2 to 1196.1]
  Anti-HPV-16, 36-45-year, Month 48: number analyzed (Participants) | 51 | 54
  Anti-HPV-16, 36-45-year, Month 48 | 2081.4 [1378.1 to 3143.6] | 1018.7 [645.3 to 1608.0]
  Anti-HPV-16, 36-45-year, Month 60: number analyzed (Participants) | 46 | 47
  Anti-HPV-16, 36-45-year, Month 60 | 1784.5 [1233.1 to 2582.6] | 764.9 [468.3 to 1249.4]
  Anti-HPV-18, 18-26-year, Month 6 | 686.2 [549.1 to 857.6] | 234.1 [186.6 to 293.5]
  Anti-HPV-18, 18-26-year, Month 12: number analyzed (Participants) | 112 | 127
  Anti-HPV-18, 18-26-year, Month 12 | 4472.4 [3528.1 to 5669.3] | 595.8 [469.0 to 756.9]
  Anti-HPV-18, 18-26-year, Month 18: number analyzed (Participants) | 109 | 114
  Anti-HPV-18, 18-26-year, Month 18 | 2256.1 [1761.5 to 2889.6] | 249.3 [195.2 to 318.3]
  Anti-HPV-18, 18-26-year, Month 24: number analyzed (Participants) | 106 | 109
  Anti-HPV-18, 18-26-year, Month 24 | 1652.0 [1296.3 to 2105.4] | 175.1 [132.8 to 230.8]
  Anti-HPV-18, 18-26-year, Month 36: number analyzed (Participants) | 64 | 76
  Anti-HPV-18, 18-26-year, Month 36 | 1593.7 [1177.2 to 2157.6] | 127.8 [92.6 to 176.6]
  Anti-HPV-18, 18-26-year, Month 48: number analyzed (Participants) | 59 | 70
  Anti-HPV-18, 18-26-year, Month 48 | 1710.9 [1179.5 to 2481.8] | 139.0 [98.7 to 195.8]
  Anti-HPV-18, 18-26-year, Month 60: number analyzed (Participants) | 39 | 52
  Anti-HPV-18, 18-26-year, Month 60 | 1522.9 [968.2 to 2395.4] | 126.2 [84.0 to 189.5]
  Anti-HPV-18, 27-35-year, Month 6: number analyzed (Participants) | 102 | 100
  Anti-HPV-18, 27-35-year, Month 6 | 429.2 [326.4 to 564.4] | 175.8 [132.8 to 232.6]
  Anti-HPV-18, 27-35-year, Month 7: number analyzed (Participants) | 110 | 102
  Anti-HPV-18, 27-35-year, Month 7 | 9501.6 [7518.5 to 12007.7] | 1043.0 [789.6 to 1377.7]
  Anti-HPV-18, 27-35-year, Month 12: number analyzed (Participants) | 105 | 102
  Anti-HPV-18, 27-35-year, Month 12 | 2266.3 [1764.8 to 2910.1] | 280.3 [209.2 to 375.5]
  Anti-HPV-18, 27-35-year, Month 18: number analyzed (Participants) | 101 | 99
  Anti-HPV-18, 27-35-year, Month 18 | 1302.2 [1011.3 to 1677.0] | 133.3 [100.8 to 176.3]
  Anti-HPV-18, 27-35-year, Month 24: number analyzed (Participants) | 98 | 94
  Anti-HPV-18, 27-35-year, Month 24 | 1028.4 [801.4 to 1319.8] | 116.2 [87.4 to 154.5]
  Anti-HPV-18, 27-35-year, Month 36: number analyzed (Participants) | 75 | 61
  Anti-HPV-18, 27-35-year, Month 36 | 942.8 [712.6 to 1247.3] | 101.9 [69.6 to 149.2]
  Anti-HPV-18, 27-35-year, Month 48: number analyzed (Participants) | 66 | 59
  Anti-HPV-18, 27-35-year, Month 48 | 982.4 [741.4 to 1301.7] | 76.9 [52.7 to 112.3]
  Anti-HPV-18, 27-35-year, Month 60: number analyzed (Participants) | 54 | 36
  Anti-HPV-18, 27-35-year, Month 60 | 967.2 [701.2 to 1334.1] | 74.4 [46.8 to 118.2]
  Anti-HPV-18, 36-45-year, Month 6: number analyzed (Participants) | 110 | 89
  Anti-HPV-18, 36-45-year, Month 6 | 618.8 [446.6 to 857.4] | 168.7 [126.9 to 224.3]
  Anti-HPV-18, 36-45-year, Month 7: number analyzed (Participants) | 110 | 91
  Anti-HPV-18, 36-45-year, Month 7 | 9845.5 [7834.7 to 12372.3] | 1438.8 [1105.0 to 1873.4]
  Anti-HPV-18, 36-45-year, Month 12: number analyzed (Participants) | 104 | 91
  Anti-HPV-18, 36-45-year, Month 12 | 3032.4 [2320.8 to 3962.3] | 433.9 [325.2 to 579.0]
  Anti-HPV-18, 36-45-year, Month 18: number analyzed (Participants) | 103 | 91
  Anti-HPV-18, 36-45-year, Month 18 | 1426.7 [1083.9 to 1877.9] | 181.5 [136.8 to 240.8]
  Anti-HPV-18, 36-45-year, Month 24: number analyzed (Participants) | 100 | 88
  Anti-HPV-18, 36-45-year, Month 24 | 1040.0 [785.7 to 1376.6] | 135.8 [99.0 to 186.2]
  Anti-HPV-18, 36-45-year, Month 36: number analyzed (Participants) | 71 | 61
  Anti-HPV-18, 36-45-year, Month 36 | 903.5 [625.1 to 1305.8] | 103.2 [74.6 to 142.8]
  Anti-HPV-18, 36-45-year, Month 48: number analyzed (Participants) | 61 | 61
  Anti-HPV-18, 36-45-year, Month 48 | 784.5 [528.7 to 1164.2] | 91.5 [67.0 to 125.0]
  Anti-HPV-18, 36-45-year, Month 60: number analyzed (Participants) | 55 | 51
  Anti-HPV-18, 36-45-year, Month 60 | 816.6 [554.7 to 1202.1] | 105.3 [71.8 to 154.3]

3. Secondary Outcome: Number of Subjects With Antibody Titers (Neutralizing Assay) Against Other Oncongenic HPV Types Greater Than or Equal to the Cut-off Value
Description: Other oncogenic HPV types include HPV-31 and HPV-45. The titer value (=serum dilution giving a 50 percent reduction of the signal compared to a control without serum) used as the cut-off for seroconversion was 40 for both other oncogenic types HPV-31 and HPV-45.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 128 | 131
Participants
  Anti-HPV-31, 18-26-year: number analyzed (Participants) | 112 | 130
  Anti-HPV-31, 18-26-year | 90 | 60
  Anti-HPV-31, 27-35-year: number analyzed (Participants) | 101 | 102
  Anti-HPV-31, 27-35-year | 59 | 32
  Anti-HPV-31, 36-45-year: number analyzed (Participants) | 102 | 99
  Anti-HPV-31, 36-45-year | 68 | 39
  Anti-HPV-45, 18-26-year | 35 | 4
  Anti-HPV-45, 27-35-year: number analyzed (Participants) | 112 | 111
  Anti-HPV-45, 27-35-year | 21 | 7
  Anti-HPV-45, 36-45-year: number analyzed (Participants) | 115 | 105
  Anti-HPV-45, 36-45-year | 28 | 10

4. Secondary Outcome: Titers of Antibodies to Other Oncogenic HPV Types Measured by Neutralization Assay
Description: Other Oncogenic Types include HPV-31 and HPV-45. Titers were measured by neutralization assay and are given as Geometric Mean Titers (GMTs). The titer is the serum dilution giving a 50 percent reduction of the signal compared to a control without serum
Time Frame: At Month 7
Population: Analysis was performed by age group on subjects from the According-to-Protocol (ATP) cohort for immunogenicity with titer greater than or equal to 40 ED50 and who were seronegative by Pseudovirion neutralizing assay and deoxyribonucleic acid (DNA) negative for the corresponding type at baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 128 | 131
titer
  Anti-HPV-31, 18-26-year: number analyzed (Participants) | 112 | 130
  Anti-HPV-31, 18-26-year | 387.3 [288.1 to 520.7] | 143.2 [110.4 to 185.8]
  Anti-HPV-31, 27-35-year: number analyzed (Participants) | 101 | 102
  Anti-HPV-31, 27-35-year | 369.6 [271.0 to 504.2] | 191.8 [122.9 to 299.5]
  Anti-HPV-31, 36-45-year: number analyzed (Participants) | 102 | 99
  Anti-HPV-31, 36-45-year | 231.0 [165.5 to 322.3] | 198.5 [142.5 to 276.6]
  Anti-HPV-45, 18-26-year | 129.7 [87.7 to 191.7] | 86.5 [11.4 to 655.1]
  Anti-HPV-45, 27-35-year: number analyzed (Participants) | 112 | 111
  Anti-HPV-45, 27-35-year | 144.1 [84.0 to 247.3] | 379.9 [90.4 to 1595.7]
  Anti-HPV-45, 36-45-year: number analyzed (Participants) | 115 | 105
  Anti-HPV-45, 36-45-year | 157.6 [103.0 to 241.1] | 79.0 [56.3 to 110.9]

5. Secondary Outcome: Number of Subjects With Antibody Titers (Neutralizing Assay) Against Human Papilloma Virus 16 (Anti-HPV-16) and Human Papilloma Virus 18 (Anti-HPV-18) Greater Than or Equal to the Cut-off Value
Description: The titer value (=serum dilution giving a 50 percent reduction of the signal compared to a control without serum) used as the cut-off for seroconversion was 40 for both HPV-16 and HPV-18.
Time Frame: At Month 6, 7, 12, 18, 24, 36, 48 and 60
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 118 | 131
Participants
  Anti-HPV-16, 18-26-year, Month 6: number analyzed (Participants) | 104 | 102
  Anti-HPV-16, 18-26-year, Month 6 | 104 | 101
  Anti-HPV-16, 18-26-year, Month 7: number analyzed (Participants) | 104 | 103
  Anti-HPV-16, 18-26-year, Month 7 | 104 | 103
  Anti-HPV-16, 18-26-year, Month 12: number analyzed (Participants) | 101 | 99
  Anti-HPV-16, 18-26-year, Month 12 | 101 | 99
  Anti-HPV-16, 18-26-year, Month 18: number analyzed (Participants) | 100 | 91
  Anti-HPV-16, 18-26-year, Month 18 | 100 | 91
  Anti-HPV-16, 18-26-year, Month 24: number analyzed (Participants) | 97 | 89
  Anti-HPV-16, 18-26-year, Month 24 | 97 | 87
  Anti-HPV-16, 18-26-year, Month 36: number analyzed (Participants) | 60 | 62
  Anti-HPV-16, 18-26-year, Month 36 | 60 | 61
  Anti-HPV-16, 18-26-year, Month 48: number analyzed (Participants) | 54 | 57
  Anti-HPV-16, 18-26-year, Month 48 | 54 | 56
  Anti-HPV-16, 18-26-year, Month 60: number analyzed (Participants) | 35 | 40
  Anti-HPV-16, 18-26-year, Month 60 | 35 | 39
  Anti-HPV-16, 27-35-year, Month 6: number analyzed (Participants) | 90 | 84
  Anti-HPV-16, 27-35-year, Month 6 | 90 | 83
  Anti-HPV-16, 27-35-year, Month 7: number analyzed (Participants) | 90 | 85
  Anti-HPV-16, 27-35-year, Month 7 | 90 | 85
  Anti-HPV-16, 27-35-year, Month 12: number analyzed (Participants) | 91 | 85
  Anti-HPV-16, 27-35-year, Month 12 | 91 | 84
  Anti-HPV-16, 27-35-year, Month 18: number analyzed (Participants) | 87 | 83
  Anti-HPV-16, 27-35-year, Month 18 | 87 | 82
  Anti-HPV-16, 27-35-year, Month 24: number analyzed (Participants) | 84 | 79
  Anti-HPV-16, 27-35-year, Month 24 | 84 | 77
  Anti-HPV-16, 27-35-year, Month 36: number analyzed (Participants) | 63 | 49
  Anti-HPV-16, 27-35-year, Month 36 | 63 | 49
  Anti-HPV-16, 27-35-year, Month 48: number analyzed (Participants) | 54 | 51
  Anti-HPV-16, 27-35-year, Month 48 | 54 | 49
  Anti-HPV-16, 27-35-year, Month 60: number analyzed (Participants) | 43 | 29
  Anti-HPV-16, 27-35-year, Month 60 | 43 | 28
  Anti-HPV-16, 36-45-year, Month 6: number analyzed (Participants) | 96 | 81
  Anti-HPV-16, 36-45-year, Month 6 | 95 | 81
  Anti-HPV-16, 36-45-year, Month 7: number analyzed (Participants) | 96 | 83
  Anti-HPV-16, 36-45-year, Month 7 | 96 | 83
  Anti-HPV-16, 36-45-year, Month 12: number analyzed (Participants) | 89 | 83
  Anti-HPV-16, 36-45-year, Month 12 | 89 | 83
  Anti-HPV-16, 36-45-year, Month 18: number analyzed (Participants) | 90 | 82
  Anti-HPV-16, 36-45-year, Month 18 | 90 | 82
  Anti-HPV-16, 36-45-year, Month 24: number analyzed (Participants) | 87 | 80
  Anti-HPV-16, 36-45-year, Month 24 | 87 | 80
  Anti-HPV-16, 36-45-year, Month 36: number analyzed (Participants) | 61 | 57
  Anti-HPV-16, 36-45-year, Month 36 | 61 | 57
  Anti-HPV-16, 36-45-year, Month 48: number analyzed (Participants) | 51 | 54
  Anti-HPV-16, 36-45-year, Month 48 | 50 | 53
  Anti-HPV-16, 36-45-year, Month 60: number analyzed (Participants) | 46 | 47
  Anti-HPV-16, 36-45-year, Month 60 | 46 | 45
  Anti-HPV-18, 18-26-year, Month 6: number analyzed (Participants) | 118 | 130
  Anti-HPV-18, 18-26-year, Month 6 | 117 | 121
  Anti-HPV-18, 18-26-year, Month 7 | 118 | 131
  Anti-HPV-18, 18-26-year, Month 12: number analyzed (Participants) | 112 | 127
  Anti-HPV-18, 18-26-year, Month 12 | 112 | 122
  Anti-HPV-18, 18-26-year, Month 18: number analyzed (Participants) | 109 | 114
  Anti-HPV-18, 18-26-year, Month 18 | 109 | 106
  Anti-HPV-18, 18-26-year, Month 24: number analyzed (Participants) | 106 | 109
  Anti-HPV-18, 18-26-year, Month 24 | 106 | 92
  Anti-HPV-18, 18-26-year, Month 36: number analyzed (Participants) | 64 | 76
  Anti-HPV-18, 18-26-year, Month 36 | 64 | 60
  Anti-HPV-18, 18-26-year, Month 48: number analyzed (Participants) | 59 | 70
  Anti-HPV-18, 18-26-year, Month 48 | 59 | 57
  Anti-HPV-18, 18-26-year, Month 60: number analyzed (Participants) | 39 | 52
  Anti-HPV-18, 18-26-year, Month 60 | 39 | 40
  Anti-HPV-18, 27-35-year, Month 6: number analyzed (Participants) | 102 | 100
  Anti-HPV-18, 27-35-year, Month 6 | 99 | 84
  Anti-HPV-18, 27-35-year, Month 7: number analyzed (Participants) | 102 | 101
  Anti-HPV-18, 27-35-year, Month 7 | 102 | 99
  Anti-HPV-18, 27-35-year, Month 12: number analyzed (Participants) | 105 | 102
  Anti-HPV-18, 27-35-year, Month 12 | 104 | 92
  Anti-HPV-18, 27-35-year, Month 18: number analyzed (Participants) | 101 | 99
  Anti-HPV-18, 27-35-year, Month 18 | 101 | 74
  Anti-HPV-18, 27-35-year, Month 24: number analyzed (Participants) | 98 | 94
  Anti-HPV-18, 27-35-year, Month 24 | 98 | 68
  Anti-HPV-18, 27-35-year, Month 36: number analyzed (Participants) | 75 | 61
  Anti-HPV-18, 27-35-year, Month 36 | 75 | 43
  Anti-HPV-18, 27-35-year, Month 48: number analyzed (Participants) | 66 | 59
  Anti-HPV-18, 27-35-year, Month 48 | 66 | 34
  Anti-HPV-18, 27-35-year, Month 60: number analyzed (Participants) | 54 | 36
  Anti-HPV-18, 27-35-year, Month 60 | 53 | 22
  Anti-HPV-18, 36-45-year, Month 6: number analyzed (Participants) | 110 | 89
  Anti-HPV-18, 36-45-year, Month 6 | 107 | 78
  Anti-HPV-18, 36-45-year, Month 7: number analyzed (Participants) | 110 | 91
  Anti-HPV-18, 36-45-year, Month 7 | 110 | 91
  Anti-HPV-18, 36-45-year, Month 12: number analyzed (Participants) | 104 | 91
  Anti-HPV-18, 36-45-year, Month 12 | 104 | 90
  Anti-HPV-18, 36-45-year, Month 18: number analyzed (Participants) | 103 | 91
  Anti-HPV-18, 36-45-year, Month 18 | 102 | 79
  Anti-HPV-18, 36-45-year, Month 24: number analyzed (Participants) | 100 | 88
  Anti-HPV-18, 36-45-year, Month 24 | 99 | 68
  Anti-HPV-18, 36-45-year, Month 36: number analyzed (Participants) | 71 | 61
  Anti-HPV-18, 36-45-year, Month 36 | 69 | 45
  Anti-HPV-18, 36-45-year, Month 48: number analyzed (Participants) | 61 | 61
  Anti-HPV-18, 36-45-year, Month 48 | 59 | 44
  Anti-HPV-18, 36-45-year, Month 60: number analyzed (Participants) | 55 | 51
  Anti-HPV-18, 36-45-year, Month 60 | 55 | 38

6. Secondary Outcome: Number of Subjects With Anti-HPV-16 and Anti-HPV-18 Immunoglobulin G (IgG) Antibody Titers Above Cut-off Values, Measured by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Cut-off values assessed were greater than or equal to 8 ELISA units per milliliter (EL.U/mL) for HPV-16 and greater than or equal to 7 EL.U/mL for HPV-18.
Time Frame: At Month 6, 7, 12, 18, 24, 36, 48 and 60
Population: Analysis was performed by age group on subjects from the ATP cohort for immunogenicity who were seronegative (by ELISA) and DNA negative for the corresponding type at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 95 | 100
Participants
  Anti-HPV-16, 18-26-year, Month 6: number analyzed (Participants) | 91 | 85
  Anti-HPV-16, 18-26-year, Month 6 | 91 | 85
  Anti-HPV-16, 18-26-year, Month 7: number analyzed (Participants) | 91 | 86
  Anti-HPV-16, 18-26-year, Month 7 | 91 | 86
  Anti-HPV-16, 18-26-year, Month 12: number analyzed (Participants) | 87 | 81
  Anti-HPV-16, 18-26-year, Month 12 | 87 | 81
  Anti-HPV-16, 18-26-year, Month 18: number analyzed (Participants) | 84 | 76
  Anti-HPV-16, 18-26-year, Month 18 | 84 | 76
  Anti-HPV-16, 18-26-year, Month 24: number analyzed (Participants) | 81 | 73
  Anti-HPV-16, 18-26-year, Month 24 | 81 | 73
  Anti-HPV-16, 18-26-year, Month 36: number analyzed (Participants) | 50 | 53
  Anti-HPV-16, 18-26-year, Month 36 | 50 | 53
  Anti-HPV-16, 18-26-year, Month 48: number analyzed (Participants) | 46 | 47
  Anti-HPV-16, 18-26-year, Month 48 | 46 | 47
  Anti-HPV-16, 18-26-year, Month 60: number analyzed (Participants) | 31 | 35
  Anti-HPV-16, 18-26-year, Month 60 | 31 | 35
  Anti-HPV-16, 27-35-year, Month 6: number analyzed (Participants) | 57 | 55
  Anti-HPV-16, 27-35-year, Month 6 | 57 | 55
  Anti-HPV-16, 27-35-year, Month 7: number analyzed (Participants) | 57 | 56
  Anti-HPV-16, 27-35-year, Month 7 | 57 | 56
  Anti-HPV-16, 27-35-year, Month 12: number analyzed (Participants) | 57 | 57
  Anti-HPV-16, 27-35-year, Month 12 | 57 | 57
  Anti-HPV-16, 27-35-year, Month 18: number analyzed (Participants) | 54 | 53
  Anti-HPV-16, 27-35-year, Month 18 | 54 | 53
  Anti-HPV-16, 27-35-year, Month 24: number analyzed (Participants) | 52 | 51
  Anti-HPV-16, 27-35-year, Month 24 | 52 | 51
  Anti-HPV-16, 27-35-year, Month 36: number analyzed (Participants) | 41 | 35
  Anti-HPV-16, 27-35-year, Month 36 | 41 | 35
  Anti-HPV-16, 27-35-year, Month 48: number analyzed (Participants) | 37 | 36
  Anti-HPV-16, 27-35-year, Month 48 | 37 | 36
  Anti-HPV-16, 27-35-year, Month 60: number analyzed (Participants) | 28 | 20
  Anti-HPV-16, 27-35-year, Month 60 | 28 | 20
  Anti-HPV-16, 36-45-year, Month 6: number analyzed (Participants) | 64 | 52
  Anti-HPV-16, 36-45-year, Month 6 | 64 | 52
  Anti-HPV-16, 36-45-year, Month 7: number analyzed (Participants) | 64 | 52
  Anti-HPV-16, 36-45-year, Month 7 | 64 | 52
  Anti-HPV-16, 36-45-year, Month 12: number analyzed (Participants) | 59 | 53
  Anti-HPV-16, 36-45-year, Month 12 | 59 | 53
  Anti-HPV-16, 36-45-year, Month 18: number analyzed (Participants) | 61 | 52
  Anti-HPV-16, 36-45-year, Month 18 | 61 | 52
  Anti-HPV-16, 36-45-year, Month 24: number analyzed (Participants) | 58 | 50
  Anti-HPV-16, 36-45-year, Month 24 | 58 | 50
  Anti-HPV-16, 36-45-year, Month 36: number analyzed (Participants) | 42 | 36
  Anti-HPV-16, 36-45-year, Month 36 | 42 | 36
  Anti-HPV-16, 36-45-year, Month 48: number analyzed (Participants) | 35 | 36
  Anti-HPV-16, 36-45-year, Month 48 | 35 | 36
  Anti-HPV-16, 36-45-year, Month 60: number analyzed (Participants) | 31 | 31
  Anti-HPV-16, 36-45-year, Month 60 | 31 | 31
  Anti-HPV-18, 18-26-year, Month 6: number analyzed (Participants) | 95 | 99
  Anti-HPV-18, 18-26-year, Month 6 | 95 | 99
  Anti-HPV-18, 18-26-year, Month 7 | 95 | 100
  Anti-HPV-18, 18-26-year, Month 12: number analyzed (Participants) | 92 | 97
  Anti-HPV-18, 18-26-year, Month 12 | 92 | 97
  Anti-HPV-18, 18-26-year, Month 18: number analyzed (Participants) | 90 | 88
  Anti-HPV-18, 18-26-year, Month 18 | 90 | 87
  Anti-HPV-18, 18-26-year, Month 24: number analyzed (Participants) | 87 | 85
  Anti-HPV-18, 18-26-year, Month 24 | 87 | 82
  Anti-HPV-18, 18-26-year, Month 36: number analyzed (Participants) | 49 | 60
  Anti-HPV-18, 18-26-year, Month 36 | 49 | 59
  Anti-HPV-18, 18-26-year, Month 48: number analyzed (Participants) | 47 | 53
  Anti-HPV-18, 18-26-year, Month 48 | 47 | 52
  Anti-HPV-18, 18-26-year, Month 60: number analyzed (Participants) | 31 | 40
  Anti-HPV-18, 18-26-year, Month 60 | 31 | 38
  Anti-HPV-18, 27-35-year, Month 6: number analyzed (Participants) | 71 | 66
  Anti-HPV-18, 27-35-year, Month 6 | 71 | 66
  Anti-HPV-18, 27-35-year, Month 7: number analyzed (Participants) | 71 | 67
  Anti-HPV-18, 27-35-year, Month 7 | 71 | 67
  Anti-HPV-18, 27-35-year, Month 12: number analyzed (Participants) | 72 | 68
  Anti-HPV-18, 27-35-year, Month 12 | 72 | 68
  Anti-HPV-18, 27-35-year, Month 18: number analyzed (Participants) | 69 | 66
  Anti-HPV-18, 27-35-year, Month 18 | 69 | 64
  Anti-HPV-18, 27-35-year, Month 24: number analyzed (Participants) | 68 | 63
  Anti-HPV-18, 27-35-year, Month 24 | 68 | 61
  Anti-HPV-18, 27-35-year, Month 36: number analyzed (Participants) | 54 | 43
  Anti-HPV-18, 27-35-year, Month 36 | 54 | 41
  Anti-HPV-18, 27-35-year, Month 48: number analyzed (Participants) | 50 | 39
  Anti-HPV-18, 27-35-year, Month 48 | 50 | 36
  Anti-HPV-18, 27-35-year, Month 60: number analyzed (Participants) | 39 | 26
  Anti-HPV-18, 27-35-year, Month 60 | 39 | 23
  Anti-HPV-18, 36-45-year, Month 6: number analyzed (Participants) | 74 | 67
  Anti-HPV-18, 36-45-year, Month 6 | 74 | 67
  Anti-HPV-18, 36-45-year, Month 7: number analyzed (Participants) | 74 | 68
  Anti-HPV-18, 36-45-year, Month 7 | 74 | 68
  Anti-HPV-18, 36-45-year, Month 12: number analyzed (Participants) | 69 | 70
  Anti-HPV-18, 36-45-year, Month 12 | 69 | 70
  Anti-HPV-18, 36-45-year, Month 18: number analyzed (Participants) | 69 | 71
  Anti-HPV-18, 36-45-year, Month 18 | 69 | 71
  Anti-HPV-18, 36-45-year, Month 24: number analyzed (Participants) | 67 | 68
  Anti-HPV-18, 36-45-year, Month 24 | 67 | 67
  Anti-HPV-18, 36-45-year, Month 36: number analyzed (Participants) | 51 | 52
  Anti-HPV-18, 36-45-year, Month 36 | 51 | 51
  Anti-HPV-18, 36-45-year, Month 48: number analyzed (Participants) | 43 | 51
  Anti-HPV-18, 36-45-year, Month 48 | 43 | 51
  Anti-HPV-18 36-45-year, Month 60: number analyzed (Participants) | 39 | 43
  Anti-HPV-18 36-45-year, Month 60 | 39 | 41

7. Secondary Outcome: Titers of Anti-HPV-16 and Anti-HPV-18 Immunoglobulin G (IgG) Antibodies Measured by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
Time Frame: At Month 6, 7, 12, 18, 24, 36, 48 and 60
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 95 | 100
EL.U/mL
  Anti-HPV-16, 18-26-year, Month 6: number analyzed (Participants) | 91 | 85
  Anti-HPV-16, 18-26-year, Month 6 | 827.7 [697.4 to 982.4] | 889.3 [710.1 to 1113.9]
  Anti-HPV-16, 18-26-year, Month 7: number analyzed (Participants) | 91 | 86
  Anti-HPV-16, 18-26-year, Month 7 | 8864.0 [7251.6 to 10834.9] | 3248.8 [2742.3 to 3848.8]
  Anti-HPV-16, 18-26-year, Month 12: number analyzed (Participants) | 87 | 81
  Anti-HPV-16, 18-26-year, Month 12 | 3332.8 [2645.1 to 4199.2] | 1137.3 [924.6 to 1398.8]
  Anti-HPV-16, 18-26-year, Month 18: number analyzed (Participants) | 84 | 76
  Anti-HPV-16, 18-26-year, Month 18 | 2266.3 [1813.2 to 2832.6] | 560.1 [434.3 to 722.3]
  Anti-HPV-16, 18-26-year, Month 24: number analyzed (Participants) | 81 | 73
  Anti-HPV-16, 18-26-year, Month 24 | 1771.9 [1424.4 to 2204.3] | 419.7 [320.6 to 549.5]
  Anti-HPV-16, 18-26-year, Month 36: number analyzed (Participants) | 50 | 53
  Anti-HPV-16, 18-26-year, Month 36 | 1373.2 [1026.0 to 1837.8] | 297.7 [214.9 to 412.3]
  Anti-HPV-16, 18-26-year, Month 48: number analyzed (Participants) | 46 | 47
  Anti-HPV-16, 18-26-year, Month 48 | 1169.1 [872.6 to 1566.4] | 247.1 [174.0 to 350.9]
  Anti-HPV-16, 18-26-year, Month 60: number analyzed (Participants) | 31 | 35
  Anti-HPV-16, 18-26-year, Month 60 | 1196.8 [830.3 to 1725.1] | 231.9 [153.7 to 349.9]
  Anti-HPV-16, 27-35-year, Month 6: number analyzed (Participants) | 57 | 55
  Anti-HPV-16, 27-35-year, Month 6 | 414.0 [313.1 to 547.4] | 715.8 [551.0 to 930.1]
  Anti-HPV-16, 27-35-year, Month 7: number analyzed (Participants) | 57 | 56
  Anti-HPV-16, 27-35-year, Month 7 | 5076.9 [3998.4 to 6446.3] | 2203.1 [1754.3 to 2766.8]
  Anti-HPV-16, 27-35-year, Month 12: number analyzed (Participants) | 57 | 57
  Anti-HPV-16, 27-35-year, Month 12 | 1978.0 [1513.8 to 2584.4] | 769.2 [596.8 to 991.4]
  Anti-HPV-16, 27-35-year, Month 18: number analyzed (Participants) | 54 | 53
  Anti-HPV-16, 27-35-year, Month 18 | 1177.3 [892.3 to 1553.3] | 384.0 [281.1 to 524.6]
  Anti-HPV-16, 27-35-year, Month 24: number analyzed (Participants) | 52 | 51
  Anti-HPV-16, 27-35-year, Month 24 | 932.8 [713.3 to 1219.8] | 300.6 [217.1 to 416.3]
  Anti-HPV-16, 27-35-year, Month 36: number analyzed (Participants) | 41 | 35
  Anti-HPV-16, 27-35-year, Month 36 | 746.3 [559.1 to 996.3] | 201.9 [141.6 to 287.9]
  Anti-HPV-16, 27-35-year, Month 48: number analyzed (Participants) | 37 | 36
  Anti-HPV-16, 27-35-year, Month 48 | 608.2 [453.8 to 815.0] | 188.7 [131.8 to 270.1]
  Anti-HPV-16, 27-35-year, Month 60: number analyzed (Participants) | 28 | 20
  Anti-HPV-16, 27-35-year, Month 60 | 602.7 [427.6 to 849.4] | 155.7 [100.4 to 241.6]
  Anti-HPV-16, 36-45-year, Month 6: number analyzed (Participants) | 64 | 52
  Anti-HPV-16, 36-45-year, Month 6 | 536.2 [401.8 to 715.5] | 690.4 [531.9 to 896.0]
  Anti-HPV-16, 36-45-year, Month 7: number analyzed (Participants) | 64 | 52
  Anti-HPV-16, 36-45-year, Month 7 | 3789.2 [2996.7 to 4791.4] | 2064.7 [1705.2 to 2500.0]
  Anti-HPV-16, 36-45-year, Month 12: number analyzed (Participants) | 59 | 53
  Anti-HPV-16, 36-45-year, Month 12 | 1521.7 [1169.1 to 1980.7] | 722.2 [586.4 to 889.6]
  Anti-HPV-16, 36-45-year, Month 18: number analyzed (Participants) | 61 | 52
  Anti-HPV-16, 36-45-year, Month 18 | 905.0 [696.9 to 1175.4] | 382.7 [294.5 to 497.4]
  Anti-HPV-16, 36-45-year, Month 24: number analyzed (Participants) | 58 | 50
  Anti-HPV-16, 36-45-year, Month 24 | 713.9 [543.9 to 936.9] | 308.4 [242.2 to 392.7]
  Anti-HPV-16, 36-45-year, Month 36: number analyzed (Participants) | 42 | 36
  Anti-HPV-16, 36-45-year, Month 36 | 540.0 [369.2 to 789.8] | 237.1 [175.0 to 321.2]
  Anti-HPV-16, 36-45-year, Month 48: number analyzed (Participants) | 35 | 36
  Anti-HPV-16, 36-45-year, Month 48 | 462.2 [311.4 to 685.8] | 225.9 [169.6 to 301.0]
  Anti-HPV-16, 36-45-year, Month 60: number analyzed (Participants) | 31 | 31
  Anti-HPV-16, 36-45-year, Month 60 | 430.3 [300.1 to 617.1] | 199.0 [145.6 to 272.0]
  Anti-HPV-18, 18-26-year, Month 6: number analyzed (Participants) | 95 | 99
  Anti-HPV-18, 18-26-year, Month 6 | 538.7 [442.6 to 655.9] | 155.4 [128.5 to 188.0]
  Anti-HPV-18, 18-26-year, Month 7 | 4246.6 [3537.2 to 5098.2] | 756.8 [625.8 to 915.2]
  Anti-HPV-18, 18-26-year, Month 12: number analyzed (Participants) | 92 | 97
  Anti-HPV-18, 18-26-year, Month 12 | 1477.9 [1189.9 to 1835.6] | 194.0 [157.3 to 239.4]
  Anti-HPV-18, 18-26-year, Month 18: number analyzed (Participants) | 90 | 88
  Anti-HPV-18, 18-26-year, Month 18 | 825.0 [650.3 to 1046.8] | 89.6 [70.1 to 114.6]
  Anti-HPV-18, 18-26-year, Month 24: number analyzed (Participants) | 87 | 85
  Anti-HPV-18, 18-26-year, Month 24 | 649.2 [512.5 to 822.5] | 70.1 [53.6 to 91.6]
  Anti-HPV-18, 18-26-year, Month 36: number analyzed (Participants) | 49 | 60
  Anti-HPV-18, 18-26-year, Month 36 | 582.1 [418.1 to 810.4] | 61.5 [44.7 to 84.7]
  Anti-HPV-18, 18-26-year, Month 48: number analyzed (Participants) | 47 | 53
  Anti-HPV-18, 18-26-year, Month 48 | 449.7 [319.0 to 633.8] | 55.1 [39.9 to 75.9]
  Anti-HPV-18, 18-26-year, Month 60: number analyzed (Participants) | 31 | 40
  Anti-HPV-18, 18-26-year, Month 60 | 451.8 [281.7 to 724.6] | 49.6 [33.0 to 74.6]
  Anti-HPV-18, 27-35-year, Month 6: number analyzed (Participants) | 71 | 66
  Anti-HPV-18, 27-35-year, Month 6 | 314.6 [245.7 to 403.0] | 128.6 [100.1 to 165.2]
  Anti-HPV-18, 27-35-year, Month 7: number analyzed (Participants) | 71 | 67
  Anti-HPV-18, 27-35-year, Month 7 | 2726.3 [2232.7 to 3329.0] | 503.4 [395.4 to 640.9]
  Anti-HPV-18, 27-35-year, Month 12: number analyzed (Participants) | 72 | 68
  Anti-HPV-18, 27-35-year, Month 12 | 892.4 [716.1 to 1112.0] | 130.4 [101.1 to 168.1]
  Anti-HPV-18, 27-35-year, Month 18: number analyzed (Participants) | 69 | 66
  Anti-HPV-18, 27-35-year, Month 18 | 501.2 [397.6 to 631.9] | 55.0 [41.8 to 72.4]
  Anti-HPV-18, 27-35-year, Month 24: number analyzed (Participants) | 68 | 63
  Anti-HPV-18, 27-35-year, Month 24 | 390.5 [311.0 to 490.4] | 46.4 [35.6 to 60.6]
  Anti-HPV-18, 27-35-year, Month 36: number analyzed (Participants) | 54 | 43
  Anti-HPV-18, 27-35-year, Month 36 | 341.7 [265.0 to 440.5] | 39.2 [27.3 to 56.2]
  Anti-HPV-18, 27-35-year, Month 48: number analyzed (Participants) | 50 | 39
  Anti-HPV-18, 27-35-year, Month 48 | 304.7 [232.4 to 399.5] | 30.6 [21.1 to 44.4]
  Anti-HPV-18, 27-35-year, Month 60: number analyzed (Participants) | 39 | 26
  Anti-HPV-18, 27-35-year, Month 60 | 231.8 [183.6 to 292.7] | 30.9 [19.0 to 50.3]
  Anti-HPV-18, 36-45-year, Month 6: number analyzed (Participants) | 74 | 67
  Anti-HPV-18, 36-45-year, Month 6 | 331.1 [253.0 to 433.2] | 131.3 [104.1 to 165.6]
  Anti-HPV-18, 36-45-year, Month 7: number analyzed (Participants) | 74 | 68
  Anti-HPV-18, 36-45-year, Month 7 | 2709.6 [2188.3 to 3355.1] | 636.2 [511.5 to 791.2]
  Anti-HPV-18, 36-45-year, Month 12: number analyzed (Participants) | 69 | 70
  Anti-HPV-18, 36-45-year, Month 12 | 838.8 [650.5 to 1081.7] | 185.0 [148.0 to 231.3]
  Anti-HPV-18, 36-45-year, Month 18: number analyzed (Participants) | 69 | 71
  Anti-HPV-18, 36-45-year, Month 18 | 454.8 [355.6 to 581.7] | 85.8 [68.8 to 107.1]
  Anti-HPV-18, 36-45-year, Month 24: number analyzed (Participants) | 67 | 68
  Anti-HPV-18, 36-45-year, Month 24 | 345.2 [266.4 to 447.2] | 66.9 [51.5 to 86.9]
  Anti-HPV-18, 36-45-year, Month 36: number analyzed (Participants) | 51 | 52
  Anti-HPV-18, 36-45-year, Month 36 | 276.8 [199.8 to 383.3] | 53.5 [40.2 to 71.3]
  Anti-HPV-18, 36-45-year, Month 48: number analyzed (Participants) | 43 | 51
  Anti-HPV-18, 36-45-year, Month 48 | 231.2 [167.9 to 318.4] | 47.8 [37.2 to 61.3]
  Anti-HPV-18, 36-45-year, Month 60: number analyzed (Participants) | 39 | 43
  Anti-HPV-18, 36-45-year, Month 60 | 242.2 [170.3 to 344.6] | 41.0 [30.5 to 55.0]

8. Secondary Outcome: Number of Subjects With Antibody Titers to Other Oncogenic HPV Types Greater Than or Equal to a Cut-off Value, Measured by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Other oncogenic types include HPV-31 and HPV-45. Cut-off values assessed were greater than or equal 59 EL.U/mL in the sera of subjects seronegative before vaccination.
Time Frame: At Month 6, 7, 12, 18, 24, 36 and 48
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 109 | 111
Participants
  Anti-HPV-31, 18-26-year, Month 6: number analyzed (Participants) | 98 | 110
  Anti-HPV-31, 18-26-year, Month 6 | 75 | 104
  Anti-HPV-31, 18-26-year, Month 7: number analyzed (Participants) | 98 | 111
  Anti-HPV-31, 18-26-year, Month 7 | 98 | 111
  Anti-HPV-31, 18-26-year, Month 12: number analyzed (Participants) | 94 | 106
  Anti-HPV-31, 18-26-year, Month 12 | 89 | 103
  Anti-HPV-31, 18-26-year, Month 18: number analyzed (Participants) | 92 | 96
  Anti-HPV-31, 18-26-year, Month 18 | 80 | 71
  Anti-HPV-31, 18-26-year, Month 24: number analyzed (Participants) | 90 | 90
  Anti-HPV-31, 18-26-year, Month 24 | 77 | 62
  Anti-HPV-31, 18-26-year, Month 36: number analyzed (Participants) | 54 | 65
  Anti-HPV-31, 18-26-year, Month 36 | 44 | 42
  Anti-HPV-31, 18-26-year, Month 48: number analyzed (Participants) | 49 | 59
  Anti-HPV-31, 18-26-year, Month 48 | 37 | 32
  Anti-HPV-31, 27-35-year, Month 6: number analyzed (Participants) | 82 | 80
  Anti-HPV-31, 27-35-year, Month 6 | 42 | 76
  Anti-HPV-31, 27-35-year, Month 7: number analyzed (Participants) | 82 | 81
  Anti-HPV-31, 27-35-year, Month 7 | 80 | 81
  Anti-HPV-31, 27-35-year, Month 12: number analyzed (Participants) | 82 | 81
  Anti-HPV-31, 27-35-year, Month 12 | 72 | 80
  Anti-HPV-31, 27-35-year, Month 18: number analyzed (Participants) | 80 | 80
  Anti-HPV-31, 27-35-year, Month 18 | 52 | 53
  Anti-HPV-31, 27-35-year, Month 24: number analyzed (Participants) | 75 | 75
  Anti-HPV-31, 27-35-year, Month 24 | 50 | 48
  Anti-HPV-31, 27-35-year, Month 36: number analyzed (Participants) | 56 | 54
  Anti-HPV-31, 27-35-year, Month 36 | 30 | 29
  Anti-HPV-31, 27-35-year, Month 48: number analyzed (Participants) | 51 | 52
  Anti-HPV-31, 27-35-year, Month 48 | 22 | 23
  Anti-HPV-31, 36-45-year, Month 6: number analyzed (Participants) | 78 | 77
  Anti-HPV-31, 36-45-year, Month 6 | 45 | 70
  Anti-HPV-31, 36-45-year, Month 7: number analyzed (Participants) | 78 | 78
  Anti-HPV-31, 36-45-year, Month 7 | 76 | 78
  Anti-HPV-31, 36-45-year, Month 18: number analyzed (Participants) | 71 | 77
  Anti-HPV-31, 36-45-year, Month 18 | 48 | 56
  Anti-HPV-31, 36-45-year, Month 12: number analyzed (Participants) | 75 | 78
  Anti-HPV-31, 36-45-year, Month 12 | 69 | 75
  Anti-HPV-31, 36-45-year, Month 24: number analyzed (Participants) | 69 | 76
  Anti-HPV-31, 36-45-year, Month 24 | 49 | 51
  Anti-HPV-31, 36-45-year, Month 36: number analyzed (Participants) | 51 | 59
  Anti-HPV-31, 36-45-year, Month 36 | 33 | 38
  Anti-HPV-31, 36-45-year, Month 48: number analyzed (Participants) | 39 | 55
  Anti-HPV-31, 36-45-year, Month 48 | 20 | 32
  Anti-HPV-45, 18-26-year, Month 6: number analyzed (Participants) | 109 | 108
  Anti-HPV-45, 18-26-year, Month 6 | 95 | 104
  Anti-HPV-45, 18-26-year, Month 7: number analyzed (Participants) | 109 | 109
  Anti-HPV-45, 18-26-year, Month 7 | 109 | 109
  Anti-HPV-45, 18-26-year, Month 12: number analyzed (Participants) | 103 | 107
  Anti-HPV-45, 18-26-year, Month 12 | 101 | 105
  Anti-HPV-45, 18-26-year, Month 18: number analyzed (Participants) | 102 | 96
  Anti-HPV-45, 18-26-year, Month 18 | 90 | 77
  Anti-HPV-45, 18-26-year, Month 24: number analyzed (Participants) | 100 | 92
  Anti-HPV-45, 18-26-year, Month 24 | 89 | 68
  Anti-HPV-45, 18-26-year, Month 36: number analyzed (Participants) | 59 | 64
  Anti-HPV-45, 18-26-year, Month 36 | 50 | 46
  Anti-HPV-45, 18-26-year, Month 48: number analyzed (Participants) | 53 | 57
  Anti-HPV-45, 18-26-year, Month 48 | 37 | 34
  Anti-HPV-45, 27-35-year, Month 6: number analyzed (Participants) | 86 | 85
  Anti-HPV-45, 27-35-year, Month 6 | 62 | 83
  Anti-HPV-45, 27-35-year, Month 7: number analyzed (Participants) | 86 | 86
  Anti-HPV-45, 27-35-year, Month 7 | 85 | 86
  Anti-HPV-45, 27-35-year, Month 12: number analyzed (Participants) | 89 | 87
  Anti-HPV-45, 27-35-year, Month 12 | 81 | 84
  Anti-HPV-45, 27-35-year, Month 18: number analyzed (Participants) | 85 | 82
  Anti-HPV-45, 27-35-year, Month 18 | 68 | 64
  Anti-HPV-45, 27-35-year, Month 24: number analyzed (Participants) | 83 | 76
  Anti-HPV-45, 27-35-year, Month 24 | 68 | 56
  Anti-HPV-45, 27-35-year, Month 36: number analyzed (Participants) | 65 | 49
  Anti-HPV-45, 27-35-year, Month 36 | 45 | 29
  Anti-HPV-45, 27-35-year, Month 48: number analyzed (Participants) | 59 | 48
  Anti-HPV-45, 27-35-year, Month 48 | 36 | 21
  Anti-HPV-45, 36-45-year, Month 6: number analyzed (Participants) | 84 | 78
  Anti-HPV-45, 36-45-year, Month 6 | 58 | 76
  Anti-HPV-45, 36-45-year, Month 7: number analyzed (Participants) | 84 | 80
  Anti-HPV-45, 36-45-year, Month 7 | 83 | 80
  Anti-HPV-45, 36-45-year, Month 12: number analyzed (Participants) | 78 | 82
  Anti-HPV-45, 36-45-year, Month 12 | 73 | 80
  Anti-HPV-45, 36-45-year, Month 18: number analyzed (Participants) | 79 | 80
  Anti-HPV-45, 36-45-year, Month 18 | 56 | 67
  Anti-HPV-45, 36-45-year, Month 24: number analyzed (Participants) | 74 | 78
  Anti-HPV-45, 36-45-year, Month 24 | 51 | 61
  Anti-HPV-45, 36-45-year, Month 36: number analyzed (Participants) | 56 | 60
  Anti-HPV-45, 36-45-year, Month 36 | 31 | 41
  Anti-HPV-45, 36-45-year, Month 48: number analyzed (Participants) | 46 | 58
  Anti-HPV-45, 36-45-year, Month 48 | 28 | 32

9. Secondary Outcome: Titers of Antibodies to Other Oncogenic HPV Types Measured by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Other oncogenic types include HPV-31 and HPV-45. Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
Time Frame: At Month 6, 7, 12, 18, 24, 36 and 48
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 109 | 111
EL.U/mL
  Anti-HPV-31, 18-26-year, Month 6: number analyzed (Participants) | 98 | 110
  Anti-HPV-31, 18-26-year, Month 6 | 108.5 [89.0 to 132.2] | 230.0 [191.7 to 276.0]
  Anti-HPV-31, 18-26-year, Month 7: number analyzed (Participants) | 98 | 111
  Anti-HPV-31, 18-26-year, Month 7 | 1245.8 [1013.0 to 1532.1] | 865.9 [734.9 to 1020.2]
  Anti-HPV-31, 18-26-year, Month 12: number analyzed (Participants) | 94 | 106
  Anti-HPV-31, 18-26-year, Month 12 | 357.0 [280.6 to 454.3] | 265.0 [221.9 to 316.4]
  Anti-HPV-31, 18-26-year, Month 18: number analyzed (Participants) | 92 | 96
  Anti-HPV-31, 18-26-year, Month 18 | 231.3 [180.8 to 295.8] | 115.1 [93.4 to 141.9]
  Anti-HPV-31, 18-26-year, Month 24: number analyzed (Participants) | 90 | 90
  Anti-HPV-31, 18-26-year, Month 24 | 214.8 [167.5 to 275.3] | 108.6 [86.0 to 137.1]
  Anti-HPV-31, 18-26-year, Month 36: number analyzed (Participants) | 54 | 65
  Anti-HPV-31, 18-26-year, Month 36 | 169.2 [125.4 to 228.3] | 94.0 [73.5 to 120.4]
  Anti-HPV-31, 18-26-year, Month 48: number analyzed (Participants) | 49 | 59
  Anti-HPV-31, 18-26-year, Month 48 | 124.7 [91.8 to 169.4] | 75.7 [58.2 to 98.4]
  Anti-HPV-31, 27-35-year, Month 6: number analyzed (Participants) | 82 | 80
  Anti-HPV-31, 27-35-year, Month 6 | 69.1 [55.1 to 86.8] | 235.9 [188.0 to 296.0]
  Anti-HPV-31, 27-35-year, Month 7: number analyzed (Participants) | 82 | 81
  Anti-HPV-31, 27-35-year, Month 7 | 588.5 [462.7 to 748.4] | 602.7 [500.0 to 726.4]
  Anti-HPV-31, 27-35-year, Month 12: number analyzed (Participants) | 82 | 81
  Anti-HPV-31, 27-35-year, Month 12 | 166.5 [130.3 to 212.8] | 217.8 [180.4 to 262.9]
  Anti-HPV-31, 27-35-year, Month 18: number analyzed (Participants) | 80 | 80
  Anti-HPV-31, 27-35-year, Month 18 | 106.0 [81.4 to 138.0] | 95.6 [75.8 to 120.7]
  Anti-HPV-31, 27-35-year, Month 24: number analyzed (Participants) | 75 | 75
  Anti-HPV-31, 27-35-year, Month 24 | 99.1 [76.7 to 128.1] | 86.7 [67.7 to 111.1]
  Anti-HPV-31, 27-35-year, Month 36: number analyzed (Participants) | 56 | 54
  Anti-HPV-31, 27-35-year, Month 36 | 74.5 [56.0 to 99.1] | 69.2 [52.4 to 91.4]
  Anti-HPV-31, 27-35-year, Month 48: number analyzed (Participants) | 51 | 52
  Anti-HPV-31, 27-35-year, Month 48 | 64.4 [48.4 to 85.8] | 59.8 [46.0 to 77.7]
  Anti-HPV-31, 36-45-year, Month 6: number analyzed (Participants) | 78 | 77
  Anti-HPV-31, 36-45-year, Month 6 | 88.4 [67.0 to 116.7] | 223.8 [169.4 to 295.6]
  Anti-HPV-31, 36-45-year, Month 7: number analyzed (Participants) | 78 | 78
  Anti-HPV-31, 36-45-year, Month 7 | 687.5 [551.2 to 857.4] | 649.6 [519.6 to 811.9]
  Anti-HPV-31, 36-45-year, Month 12: number analyzed (Participants) | 75 | 78
  Anti-HPV-31, 36-45-year, Month 12 | 197.1 [154.5 to 251.5] | 243.5 [191.6 to 309.4]
  Anti-HPV-31, 36-45-year, Month 18: number analyzed (Participants) | 71 | 77
  Anti-HPV-31, 36-45-year, Month 18 | 109.5 [83.1 to 144.4] | 122.9 [93.2 to 162.1]
  Anti-HPV-31, 36-45-year, Month 24: number analyzed (Participants) | 69 | 76
  Anti-HPV-31, 36-45-year, Month 24 | 108.8 [83.5 to 141.7] | 110.6 [83.2 to 147.0]
  Anti-HPV-31, 36-45-year, Month 36: number analyzed (Participants) | 51 | 59
  Anti-HPV-31, 36-45-year, Month 36 | 94.4 [69.6 to 128.1] | 92.8 [69.5 to 124.0]
  Anti-HPV-31, 36-45-year, Month 48: number analyzed (Participants) | 39 | 55
  Anti-HPV-31, 36-45-year, Month 48 | 67.4 [49.3 to 92.1] | 71.8 [54.8 to 94.0]
  Anti-HPV-45, 18-26-year, Month 6: number analyzed (Participants) | 109 | 108
  Anti-HPV-45, 18-26-year, Month 6 | 155.4 [130.2 to 185.5] | 242.6 [203.3 to 289.6]
  Anti-HPV-45, 18-26-year, Month 7: number analyzed (Participants) | 109 | 109
  Anti-HPV-45, 18-26-year, Month 7 | 1248.1 [1040.8 to 1496.6] | 1103.5 [938.9 to 1296.9]
  Anti-HPV-45, 18-26-year, Month 12: number analyzed (Participants) | 103 | 107
  Anti-HPV-45, 18-26-year, Month 12 | 348.0 [283.2 to 427.7] | 277.8 [235.3 to 328.0]
  Anti-HPV-45, 18-26-year, Month 18: number analyzed (Participants) | 102 | 96
  Anti-HPV-45, 18-26-year, Month 18 | 216.2 [170.6 to 273.9] | 127.1 [103.6 to 155.9]
  Anti-HPV-45, 18-26-year, Month 24: number analyzed (Participants) | 100 | 92
  Anti-HPV-45, 18-26-year, Month 24 | 192.9 [154.4 to 240.8] | 114.0 [91.7 to 141.7]
  Anti-HPV-45, 18-26-year, Month 36: number analyzed (Participants) | 59 | 64
  Anti-HPV-45, 18-26-year, Month 36 | 140.5 [106.7 to 184.9] | 95.2 [76.5 to 118.6]
  Anti-HPV-45, 18-26-year, Month 48: number analyzed (Participants) | 53 | 57
  Anti-HPV-45, 18-26-year, Month 48 | 99.8 [74.3 to 134.0] | 75.6 [57.6 to 99.4]
  Anti-HPV-45, 27-35-year, Month 6: number analyzed (Participants) | 86 | 85
  Anti-HPV-45, 27-35-year, Month 6 | 103.3 [82.1 to 130.0] | 260.7 [212.4 to 319.9]
  Anti-HPV-45, 27-35-year, Month 7: number analyzed (Participants) | 86 | 86
  Anti-HPV-45, 27-35-year, Month 7 | 720.6 [579.2 to 896.6] | 828.8 [695.6 to 987.3]
  Anti-HPV-45, 27-35-year, Month 12: number analyzed (Participants) | 89 | 87
  Anti-HPV-45, 27-35-year, Month 12 | 212.1 [168.9 to 266.3] | 242.3 [201.2 to 291.8]
  Anti-HPV-45, 27-35-year, Month 18: number analyzed (Participants) | 85 | 82
  Anti-HPV-45, 27-35-year, Month 18 | 135.3 [106.5 to 171.9] | 102.0 [84.0 to 123.9]
  Anti-HPV-45, 27-35-year, Month 24: number analyzed (Participants) | 83 | 76
  Anti-HPV-45, 27-35-year, Month 24 | 125.9 [101.3 to 156.5] | 100.6 [79.1 to 127.9]
  Anti-HPV-45, 27-35-year, Month 36: number analyzed (Participants) | 65 | 49
  Anti-HPV-45, 27-35-year, Month 36 | 94.3 [73.9 to 120.5] | 73.5 [56.0 to 96.5]
  Anti-HPV-45, 27-35-year, Month 48: number analyzed (Participants) | 59 | 48
  Anti-HPV-45, 27-35-year, Month 48 | 79.1 [61.3 to 102.0] | 60.2 [45.9 to 78.9]
  Anti-HPV-45, 36-45-year, Month 6: number analyzed (Participants) | 84 | 78
  Anti-HPV-45, 36-45-year, Month 6 | 103.0 [80.8 to 131.4] | 258.8 [204.7 to 327.3]
  Anti-HPV-45, 36-45-year, Month 7: number analyzed (Participants) | 84 | 80
  Anti-HPV-45, 36-45-year, Month 7 | 634.3 [506.1 to 795.0] | 985.1 [803.8 to 1207.4]
  Anti-HPV-45, 36-45-year, Month 12: number analyzed (Participants) | 78 | 82
  Anti-HPV-45, 36-45-year, Month 12 | 196.3 [154.8 to 248.8] | 298.2 [243.1 to 365.8]
  Anti-HPV-45, 36-45-year, Month 18: number analyzed (Participants) | 79 | 80
  Anti-HPV-45, 36-45-year, Month 18 | 121.7 [93.5 to 158.5] | 141.6 [113.3 to 177.0]
  Anti-HPV-45, 36-45-year, Month 24: number analyzed (Participants) | 74 | 78
  Anti-HPV-45, 36-45-year, Month 24 | 114.1 [87.6 to 148.8] | 122.7 [97.2 to 155.0]
  Anti-HPV-45, 36-45-year, Month 36: number analyzed (Participants) | 56 | 60
  Anti-HPV-45, 36-45-year, Month 36 | 85.5 [63.9 to 114.5] | 94.7 [73.6 to 121.8]
  Anti-HPV-45, 36-45-year, Month 48: number analyzed (Participants) | 46 | 58
  Anti-HPV-45, 36-45-year, Month 48 | 82.8 [61.8 to 111.0] | 74.3 [57.8 to 95.5]

10. Secondary Outcome: Number of HPV-16 and HVP-18 Specific CD4 Cells Producing at Least 2 Different Cytokines Per Million of CD4 T Cells
Description: Number of cells were expressed as geometric mean, minimum and maximum values of specific CD4 cells producing at least 2 cytokines (CD40 Ligand, Interleukin-2, Tumor Necrosis Factor Alpha or Interferon-gamma) per million of CD4 T-cells.
Time Frame: At Month 7, 12, 18, 24, 36 and 48
Population: Results are presented by age group for subjects HPV-16/18 seronegative (by PSV neutralizing assay), DNA negative and HPV-16/18 specific T-cell negative (i.e., with < 500 cells/million cells at baseline) from a subset of the ATP cohort for immunogenicity.
Measure: Geometric Mean (Full Range); unit: cells per million CD4 T-cells
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 17 | 18
cells per million CD4 T-cells
  HPV-16, 18-26-year, Month 7: number analyzed (Participants) | 12 | 13
  HPV-16, 18-26-year, Month 7 | 1285.6 [695.0 to 3040.0] | 729.1 [277.0 to 2515.0]
  HPV-16, 18-26-year, Month 12: number analyzed (Participants) | 10 | 9
  HPV-16, 18-26-year, Month 12 | 1087.6 [400.0 to 3203.0] | 421.3 [187.0 to 1239.0]
  HPV-16, 18-26-year, Month 18: number analyzed (Participants) | 14 | 8
  HPV-16, 18-26-year, Month 18 | 1194.4 [508.0 to 3902.0] | 309.0 [26.0 to 1281.0]
  HPV-16, 18-26-year, Month 24: number analyzed (Participants) | 13 | 8
  HPV-16, 18-26-year, Month 24 | 1195.9 [632.0 to 2979.0] | 323.5 [72.0 to 919.0]
  HPV-16, 18-26-year, Month 36: number analyzed (Participants) | 6 | 6
  HPV-16, 18-26-year, Month 36 | 838.3 [379.0 to 1309.0] | 399.9 [175.0 to 789.0]
  HPV-16, 18-26-year, Month 48: number analyzed (Participants) | 3 | 6
  HPV-16, 18-26-year, Month 48 | 1272.4 [994.0 to 1658.0] | 388.6 [208.0 to 958.0]
  HPV-16, 27-35-year, Month 7: number analyzed (Participants) | 15 | 12
  HPV-16, 27-35-year, Month 7 | 990.7 [54.0 to 4231.0] | 637.1 [172.0 to 1990.0]
  HPV-16, 27-35-year, Month 12: number analyzed (Participants) | 13 | 9
  HPV-16, 27-35-year, Month 12 | 664.1 [112.0 to 1762.0] | 493.3 [227.0 to 1230.0]
  HPV-16, 27-35-year, Month 18: number analyzed (Participants) | 13 | 8
  HPV-16, 27-35-year, Month 18 | 1134.4 [425.0 to 2158.0] | 448.0 [127.0 to 1478.0]
  HPV-16, 27-35-year, Month 24: number analyzed (Participants) | 12 | 6
  HPV-16, 27-35-year, Month 24 | 919.8 [120.0 to 2341.0] | 373.0 [81.0 to 853.0]
  HPV-16, 27-35-year, Month 36: number analyzed (Participants) | 7 | 4
  HPV-16, 27-35-year, Month 36 | 431.0 [1.0 to 2912.0] | 85.9 [1.0 to 607.0]
  HPV-16, 27-35-year, Month 48: number analyzed (Participants) | 5 | 4
  HPV-16, 27-35-year, Month 48 | 307.7 [1.0 to 1930.0] | 560.8 [285.0 to 1482.0]
  HPV-16, 36-45-year, Month 7: number analyzed (Participants) | 13 | 8
  HPV-16, 36-45-year, Month 7 | 979.7 [227.0 to 2773.0] | 609.8 [347.0 to 1320.0]
  HPV-16, 36-45-year, Month 12: number analyzed (Participants) | 10 | 9
  HPV-16, 36-45-year, Month 12 | 707.7 [200.0 to 1495.0] | 431.3 [120.0 to 936.0]
  HPV-16, 36-45-year, Month 18: number analyzed (Participants) | 13 | 9
  HPV-16, 36-45-year, Month 18 | 1116.8 [266.0 to 2840.0] | 446.1 [41.0 to 1610.0]
  HPV-16, 36-45-year, Month 24: number analyzed (Participants) | 8 | 6
  HPV-16, 36-45-year, Month 24 | 1118.9 [447.0 to 1940.0] | 789.3 [570.0 to 1090.0]
  HPV-16, 36-45-year, Month 36: number analyzed (Participants) | 7 | 5
  HPV-16, 36-45-year, Month 36 | 710.5 [71.0 to 1698.0] | 494.2 [336.0 to 1105.0]
  HPV-16, 36-45-year, Month 48: number analyzed (Participants) | 5 | 4
  HPV-16, 36-45-year, Month 48 | 1247.9 [597.0 to 2503.0] | 642.4 [367.0 to 1422.0]
  HPV-18, 18-26-year, Month 7: number analyzed (Participants) | 11 | 18
  HPV-18, 18-26-year, Month 7 | 998.8 [439.0 to 2344.0] | 594.9 [122.0 to 1783.0]
  HPV-18, 18-26-year, Month 12: number analyzed (Participants) | 8 | 13
  HPV-18, 18-26-year, Month 12 | 716.4 [238.0 to 1413.0] | 192.3 [1.0 to 906.0]
  HPV-18, 18-26-year, Month 18: number analyzed (Participants) | 13 | 13
  HPV-18, 18-26-year, Month 18 | 844.3 [346.0 to 2492.0] | 264.2 [1.0 to 1214.0]
  HPV-18, 18-26-year, Month 24: number analyzed (Participants) | 11 | 12
  HPV-18, 18-26-year, Month 24 | 793.0 [296.0 to 2051.0] | 197.4 [1.0 to 625.0]
  HPV-18, 18-26-year, Month 36: number analyzed (Participants) | 5 | 9
  HPV-18, 18-26-year, Month 36 | 622.6 [311.0 to 920.0] | 211.4 [68.0 to 557.0]
  HPV-18, 18-26-year, Month 48: number analyzed (Participants) | 3 | 9
  HPV-18, 18-26-year, Month 48 | 927.7 [819.0 to 1055.0] | 162.1 [13.0 to 676.0]
  HPV-18, 27-35-year, Month 7: number analyzed (Participants) | 17 | 14
  HPV-18, 27-35-year, Month 7 | 924.3 [217.0 to 2589.0] | 680.7 [133.0 to 2427.0]
  HPV-18, 27-35-year, Month 12: number analyzed (Participants) | 16 | 11
  HPV-18, 27-35-year, Month 12 | 416.5 [1.0 to 2239.0] | 471.2 [133.0 to 1134.0]
  HPV-18, 27-35-year, Month 18: number analyzed (Participants) | 14 | 11
  HPV-18, 27-35-year, Month 18 | 710.8 [102.0 to 1879.0] | 568.4 [106.0 to 1919.0]
  HPV-18, 27-35-year, Month 24: number analyzed (Participants) | 15 | 7
  HPV-18, 27-35-year, Month 24 | 575.6 [67.0 to 2113.0] | 355.8 [114.0 to 826.0]
  HPV-18, 27-35-year, Month 36: number analyzed (Participants) | 9 | 4
  HPV-18, 27-35-year, Month 36 | 265.4 [1.0 to 1646.0] | 206.2 [27.0 to 748.0]
  HPV-18, 27-35-year, Month 48: number analyzed (Participants) | 6 | 3
  HPV-18, 27-35-year, Month 48 | 643.7 [119.0 to 2032.0] | 426.7 [242.0 to 1198.0]
  HPV-18, 36-45-year, Month 7: number analyzed (Participants) | 14 | 8
  HPV-18, 36-45-year, Month 7 | 815.6 [147.0 to 2983.0] | 212.2 [1.0 to 1424.0]
  HPV-18, 36-45-year, Month 12: number analyzed (Participants) | 13 | 8
  HPV-18, 36-45-year, Month 12 | 384.3 [1.0 to 1521.0] | 405.0 [123.0 to 1044.0]
  HPV-18, 36-45-year, Month 18: number analyzed (Participants) | 14 | 9
  HPV-18, 36-45-year, Month 18 | 949.0 [106.0 to 2746.0] | 195.4 [1.0 to 1204.0]
  HPV-18, 36-45-year, Month 24: number analyzed (Participants) | 9 | 6
  HPV-18, 36-45-year, Month 24 | 807.2 [327.0 to 1616.0] | 520.5 [220.0 to 717.0]
  HPV-18, 36-45-year, Month 36: number analyzed (Participants) | 8 | 4
  HPV-18, 36-45-year, Month 36 | 337.4 [7.0 to 1293.0] | 392.1 [203.0 to 772.0]
  HPV-18, 36-45-year, Month 48: number analyzed (Participants) | 5 | 3
  HPV-18, 36-45-year, Month 48 | 764.0 [231.0 to 2068.0] | 612.2 [389.0 to 778.0]

11. Secondary Outcome: Number of HPV-16 and HVP-18 Specific CD8 Cells Producing at Least 2 Different Cytokines Per Million of CD8 T Cells
Description: Data were expressed as geometric mean, minimum and maximum values of specific CD8 cells producing at least 2 cytokines (CD40 Ligand, Interleukin-2, Tumor Necrosis Factor Alpha or Interferon-gamma) per million of CD8 T-cells.
  Analyses for further time points were not performed, as there was no response at these time points.
Time Frame: At Month 7, 12 and 18
Population: Results are presented by age group for subjects HPV-16/18 seronegative (by PSV neutralizing assay), DNA negative and HPV-16/18 specific T-cell negative (i.e., with < 200 cells/million cells at baseline) from a subset of the ATP cohort for immunogenicity.
Measure: Geometric Mean (Full Range); unit: cells per million CD8 T-cells
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 24 | 23
cells per million CD8 T-cells
  HPV-16, 18-26-year, Month 7: number analyzed (Participants) | 15 | 21
  HPV-16, 18-26-year, Month 7 | 5.3 [1.0 to 258.0] | 3.2 [1.0 to 107.0]
  HPV-16, 18-26-year, Month 12: number analyzed (Participants) | 17 | 21
  HPV-16, 18-26-year, Month 12 | 4.0 [1.0 to 96.0] | 2.8 [1.0 to 102.0]
  HPV-16, 18-26-year, Month 18: number analyzed (Participants) | 23 | 22
  HPV-16, 18-26-year, Month 18 | 3.5 [1.0 to 336.0] | 4.5 [1.0 to 73.0]
  HPV-16, 27-35-year, Month 7: number analyzed (Participants) | 21 | 23
  HPV-16, 27-35-year, Month 7 | 2.5 [1.0 to 89.0] | 5.1 [1.0 to 302.0]
  HPV-16, 27-35-year, Month 12: number analyzed (Participants) | 22 | 18
  HPV-16, 27-35-year, Month 12 | 5.0 [1.0 to 133.0] | 3.8 [1.0 to 205.0]
  HPV-16, 27-35-year, Month 18: number analyzed (Participants) | 22 | 20
  HPV-16, 27-35-year, Month 18 | 2.4 [1.0 to 76.0] | 8.6 [1.0 to 112.0]
  HPV-16, 36-45-year, Month 7: number analyzed (Participants) | 23 | 14
  HPV-16, 36-45-year, Month 7 | 3.0 [1.0 to 422.0] | 6.1 [1.0 to 222.0]
  HPV-16, 36-45-year, Month 12: number analyzed (Participants) | 19 | 22
  HPV-16, 36-45-year, Month 12 | 4.6 [1.0 to 123.0] | 4.0 [1.0 to 247.0]
  HPV-16, 36-45-year, Month 18: number analyzed (Participants) | 24 | 18
  HPV-16, 36-45-year, Month 18 | 4.1 [1.0 to 111.0] | 8.9 [1.0 to 412.0]
  HPV-18, 18-26-year, Month 7: number analyzed (Participants) | 16 | 20
  HPV-18, 18-26-year, Month 7 | 9.3 [1.0 to 148.0] | 3.0 [1.0 to 426.0]
  HPV-18, 18-26-year, Month 12: number analyzed (Participants) | 17 | 21
  HPV-18, 18-26-year, Month 12 | 4.6 [1.0 to 197.0] | 3.4 [1.0 to 104.0]
  HPV-18, 18-26-year, Month 18: number analyzed (Participants) | 23 | 22
  HPV-18, 18-26-year, Month 18 | 4.1 [1.0 to 533.0] | 4.3 [1.0 to 94.0]
  HPV-18, 27-35-year, Month 7: number analyzed (Participants) | 21 | 23
  HPV-18, 27-35-year, Month 7 | 2.6 [1.0 to 131.0] | 3.6 [1.0 to 173.0]
  HPV-18, 27-35-year, Month 12: number analyzed (Participants) | 22 | 18
  HPV-18, 27-35-year, Month 12 | 3.5 [1.0 to 251.0] | 4.6 [1.0 to 78.0]
  HPV-18, 27-35-year, Month 18: number analyzed (Participants) | 22 | 20
  HPV-18, 27-35-year, Month 18 | 3.1 [1.0 to 476.0] | 7.1 [1.0 to 790.0]
  HPV-18, 36-45-year, Month 7: number analyzed (Participants) | 22 | 14
  HPV-18, 36-45-year, Month 7 | 9.2 [1.0 to 202.0] | 3.4 [1.0 to 220.0]
  HPV-18, 36-45-year, Month 12: number analyzed (Participants) | 19 | 20
  HPV-18, 36-45-year, Month 12 | 2.4 [1.0 to 111.0] | 6.8 [1.0 to 261.0]
  HPV-18, 36-45-year, Month 18: number analyzed (Participants) | 23 | 18
  HPV-18, 36-45-year, Month 18 | 6.3 [1.0 to 161.0] | 4.5 [1.0 to 668.0]

12. Secondary Outcome: Number of HPV-16 and HVP-18 Specific B-cells Per Million B Cells
Description: HPV-16 and HPV-18 Specific Memory B Cells were measured by Enzyme-linked immunosorbent spot (ELISPOT) assay and expressed as geometric mean, minimum and maximum values of specific B-cells per million of cells.
Time Frame: At Month 7, 12, 18, 24, 36 and 48
Population: Results are presented by age group in subjects with detectable B-cells (>0) at defined time points, who were HPV-16/18 seronegative (by PSV neutralizing assay), DNA negative and HPV-16/18 specific B-cell negative at baseline from a subset of the ATP cohort for immunogenicity.
Measure: Geometric Mean (Full Range); unit: cells per million B-cells
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 19 | 15
cells per million B-cells
  HPV-16, 18-26-year, Month 7: number analyzed (Participants) | 13 | 13
  HPV-16, 18-26-year, Month 7 | 700.7 [223.0 to 3515.0] | 358.5 [22.0 to 2802.0]
  HPV-16, 18-26-year, Month 12: number analyzed (Participants) | 12 | 6
  HPV-16, 18-26-year, Month 12 | 344.1 [93.0 to 1068.0] | 192.3 [77.0 to 463.0]
  HPV-16, 18-26-year, Month 18: number analyzed (Participants) | 13 | 5
  HPV-16, 18-26-year, Month 18 | 262.1 [51.0 to 1067.0] | 325.2 [35.0 to 1868.0]
  HPV-16, 18-26-year, Month 24: number analyzed (Participants) | 10 | 4
  HPV-16, 18-26-year, Month 24 | 233.5 [59.0 to 1777.0] | 440.0 [30.0 to 1751.0]
  HPV-16, 18-26-year, Month 36: number analyzed (Participants) | 4 | 2
  HPV-16, 18-26-year, Month 36 | 207.7 [39.0 to 586.0] | 505.4 [445.0 to 574.0]
  HPV-16, 18-26-year, Month 48: number analyzed (Participants) | 3 | 3
  HPV-16, 18-26-year, Month 48 | 219.7 [60.0 to 657.0] | 130.0 [54.0 to 515.0]
  HPV-16, 27-35-year, Month 7: number analyzed (Participants) | 17 | 15
  HPV-16, 27-35-year, Month 7 | 898.0 [111.0 to 5058.0] | 253.5 [62.0 to 767.0]
  HPV-16, 27-35-year, Month 12: number analyzed (Participants) | 15 | 12
  HPV-16, 27-35-year, Month 12 | 237.6 [27.0 to 2910.0] | 202.8 [38.0 to 655.0]
  HPV-16, 27-35-year, Month 18: number analyzed (Participants) | 14 | 7
  HPV-16, 27-35-year, Month 18 | 216.5 [47.0 to 1846.0] | 194.3 [94.0 to 816.0]
  HPV-16, 27-35-year, Month 24: number analyzed (Participants) | 11 | 8
  HPV-16, 27-35-year, Month 24 | 279.1 [49.0 to 962.0] | 141.2 [29.0 to 715.0]
  HPV-16, 27-35-year, Month 36: number analyzed (Participants) | 4 | 6
  HPV-16, 27-35-year, Month 36 | 506.5 [270.0 to 1438.0] | 142.1 [43.0 to 290.0]
  HPV-16, 27-35-year, Month 48: number analyzed (Participants) | 4 | 3
  HPV-16, 27-35-year, Month 48 | 354.3 [72.0 to 3847.0] | 358.0 [251.0 to 456.0]
  HPV-16, 36-45-year, Month 7: number analyzed (Participants) | 15 | 7
  HPV-16, 36-45-year, Month 7 | 1476.0 [349.0 to 19927.0] | 539.3 [114.0 to 7359.0]
  HPV-16, 36-45-year, Month 12: number analyzed (Participants) | 13 | 7
  HPV-16, 36-45-year, Month 12 | 363.7 [69.0 to 1549.0] | 270.8 [37.0 to 2238.0]
  HPV-16, 36-45-year, Month 18: number analyzed (Participants) | 12 | 5
  HPV-16, 36-45-year, Month 18 | 301.3 [43.0 to 2053.0] | 210.2 [156.0 to 264.0]
  HPV-16, 36-45-year, Month 24: number analyzed (Participants) | 9 | 4
  HPV-16, 36-45-year, Month 24 | 492.1 [133.0 to 1708.0] | 338.0 [77.0 to 808.0]
  HPV-16, 36-45-year, Month 36: number analyzed (Participants) | 3 | 3
  HPV-16, 36-45-year, Month 36 | 503.9 [190.0 to 1052.0] | 192.9 [118.0 to 468.0]
  HPV-16, 36-45-year, Month 48: number analyzed (Participants) | 3 | 1
  HPV-16, 36-45-year, Month 48 | 364.8 [127.0 to 741.0] | 738.0 [738.0 to 738.0]
  HPV-18, 18-26-year, Month 7: number analyzed (Participants) | 10 | 14
  HPV-18, 18-26-year, Month 7 | 313.2 [41.0 to 792.0] | 163.9 [22.0 to 630.0]
  HPV-18, 18-26-year, Month 12: number analyzed (Participants) | 10 | 6
  HPV-18, 18-26-year, Month 12 | 152.5 [30.0 to 918.0] | 63.8 [28.0 to 181.0]
  HPV-18, 18-26-year, Month 18: number analyzed (Participants) | 10 | 8
  HPV-18, 18-26-year, Month 18 | 137.3 [31.0 to 1677.0] | 76.4 [19.0 to 479.0]
  HPV-18, 18-26-year, Month 24: number analyzed (Participants) | 9 | 9
  HPV-18, 18-26-year, Month 24 | 255.5 [36.0 to 1456.0] | 101.0 [34.0 to 668.0]
  HPV-18, 18-26-year, Month 36: number analyzed (Participants) | 3 | 3
  HPV-18, 18-26-year, Month 36 | 391.0 [87.0 to 2781.0] | 114.1 [36.0 to 779.0]
  HPV-18, 18-26-year, Month 48: number analyzed (Participants) | 3 | 4
  HPV-18, 18-26-year, Month 48 | 124.7 [46.0 to 214.0] | 118.0 [46.0 to 347.0]
  HPV-18, 27-35-year, Month 7: number analyzed (Participants) | 18 | 10
  HPV-18, 27-35-year, Month 7 | 433.4 [32.0 to 3375.0] | 153.7 [42.0 to 530.0]
  HPV-18, 27-35-year, Month 12: number analyzed (Participants) | 15 | 7
  HPV-18, 27-35-year, Month 12 | 172.4 [10.0 to 972.0] | 130.4 [20.0 to 409.0]
  HPV-18, 27-35-year, Month 18: number analyzed (Participants) | 13 | 6
  HPV-18, 27-35-year, Month 18 | 202.5 [28.0 to 869.0] | 74.7 [15.0 to 710.0]
  HPV-18, 27-35-year, Month 24: number analyzed (Participants) | 12 | 4
  HPV-18, 27-35-year, Month 24 | 151.6 [14.0 to 606.0] | 97.0 [45.0 to 226.0]
  HPV-18, 27-35-year, Month 36: number analyzed (Participants) | 5 | 4
  HPV-18, 27-35-year, Month 36 | 161.9 [53.0 to 629.0] | 224.2 [47.0 to 829.0]
  HPV-18, 27-35-year, Month 48: number analyzed (Participants) | 5 | 3
  HPV-18, 27-35-year, Month 48 | 366.4 [13.0 to 2167.0] | 134.2 [104.0 to 157.0]
  HPV-18, 36-45-year, Month 7: number analyzed (Participants) | 19 | 7
  HPV-18, 36-45-year, Month 7 | 785.7 [85.0 to 7635.0] | 192.5 [76.0 to 517.0]
  HPV-18, 36-45-year, Month 12: number analyzed (Participants) | 12 | 4
  HPV-18, 36-45-year, Month 12 | 459.8 [110.0 to 2653.0] | 242.8 [116.0 to 664.0]
  HPV-18, 36-45-year, Month 18: number analyzed (Participants) | 12 | 5
  HPV-18, 36-45-year, Month 18 | 436.9 [93.0 to 1753.0] | 91.5 [23.0 to 349.0]
  HPV-18, 36-45-year, Month 24: number analyzed (Participants) | 8 | 5
  HPV-18, 36-45-year, Month 24 | 576.8 [154.0 to 1873.0] | 106.6 [61.0 to 171.0]
  HPV-18, 36-45-year, Month 36: number analyzed (Participants) | 4 | 1
  HPV-18, 36-45-year, Month 36 | 376.6 [95.0 to 1161.0] | 23.0 [23.0 to 23.0]
  HPV-18, 36-45-year, Month 48: number analyzed (Participants) | 3 | 2
  HPV-18, 36-45-year, Month 48 | 302.4 [190.0 to 543.0] | 91.7 [69.0 to 122.0]

13. Secondary Outcome: Titers of HPV-16 IgG and HPV-18 IgG (by ELISA) in Cervico-vaginal Secretions (CVS)
Description: as for outcome 7
Time Frame: At Month 7, 12, 18, 24, 36 and 48
Population: Analyses were done on those subjects from the ATP cohort for immunogenicity for whom CVS samples with less than 200 erythrocytes per microliter were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Groups:
- Cervarix Group: Subjects received 3 doses of GSK Biologicals HPV 16/18 vaccine 580299 (CervarixTM) at Months 0, 1 and 6 and a dose of placebo at Month 2. All doses were administered by intramuscular injection in the deltoid muscle of the upper arm.
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 51 | 57
EL.U/mL
  Anti-HPV-16, Month 7: number analyzed (Participants) | 48 | 57
  Anti-HPV-16, Month 7 | 168.9 [114.4 to 249.4] | 90.7 [62.6 to 131.6]
  Anti-HPV-16, Month 12: number analyzed (Participants) | 51 | 46
  Anti-HPV-16, Month 12 | 129.7 [89.6 to 187.8] | 46.8 [33.0 to 66.5]
  Anti-HPV-16, Month 18: number analyzed (Participants) | 42 | 43
  Anti-HPV-16, Month 18 | 96.0 [64.8 to 142.3] | 52.8 [35.6 to 78.3]
  Anti-HPV-16, Month 24: number analyzed (Participants) | 45 | 43
  Anti-HPV-16, Month 24 | 85.0 [57.9 to 124.8] | 45.1 [27.0 to 75.2]
  Anti-HPV-16, Month 36: number analyzed (Participants) | 50 | 44
  Anti-HPV-16, Month 36 | 57.1 [39.6 to 82.4] | 48.8 [30.8 to 77.4]
  Anti-HPV-16, Month 48: number analyzed (Participants) | 31 | 36
  Anti-HPV-16, Month 48 | 32.7 [22.7 to 47.1] | 72.2 [34.4 to 151.3]
  Anti-HPV-18, Month 7: number analyzed (Participants) | 48 | 57
  Anti-HPV-18, Month 7 | 88.6 [65.0 to 120.8] | 43.4 [30.1 to 62.6]
  Anti-HPV-18, Month 12: number analyzed (Participants) | 51 | 47
  Anti-HPV-18, Month 12 | 59.0 [42.5 to 81.9] | 29.1 [18.6 to 45.3]
  Anti-HPV-18, Month 18: number analyzed (Participants) | 42 | 43
  Anti-HPV-18, Month 18 | 33.2 [21.3 to 51.8] | 16.4 [10.4 to 25.9]
  Anti-HPV-18, Month 24: number analyzed (Participants) | 45 | 43
  Anti-HPV-18, Month 24 | 43.9 [28.1 to 68.8] | 21.5 [10.5 to 44.3]
  Anti-HPV-18, Month 36: number analyzed (Participants) | 50 | 44
  Anti-HPV-18, Month 36 | 24.3 [18.0 to 32.8] | 23.3 [12.3 to 44.0]
  Anti-HPV-18, Month 48: number analyzed (Participants) | 31 | 36
  Anti-HPV-18, Month 48 | 16.6 [10.3 to 26.7] | 20.2 [12.5 to 32.8]

14. Secondary Outcome: Number of Subjects Completing the 3-dose Vaccination Schedule
Time Frame: Up to Month 7
Population: The number of subjects completing the 3-dose vaccination schedule was defined as the number of subjects who received the 3 active doses (placebo administrations are not reflected).
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants | 468 | 467

15. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site. All solicited local symptoms were assessed as related to study vaccination.
Time Frame: During the 7-day period (Day 0-6) following vaccination
Population: Analyses were performed on subjects with available data within the Total Vaccinated cohort, which included subjects with at least one vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 524 | 524
Participants
  Any Pain | 487 | 375
  Any Redness | 232 | 134
  Any Swelling | 191 | 114
  Grade 3 Pain | 91 | 18
  Grade 3 Redness | 3 | 0
  Grade 3 Swelling | 5 | 3

16. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], gastrointestinal, headache, myalgia, rash and urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day period (Day 0-6) following vaccination
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 526 | 525
Participants
  Any Arthralgia | 114 | 81
  Any Fatigue | 262 | 209
  Any Fever | 76 | 58
  Any Gastrointestinal symptoms | 172 | 139
  Any Headache | 250 | 220
  Any Myalgia | 145 | 103
  Any Rash | 25 | 18
  Any Urticaria | 26 | 21
  Grade 3 Arthralgia | 13 | 3
  Grade 3 Fatigue | 30 | 12
  Grade 3 Fever | 2 | 0
  Grade 3 Gastrointestinal symptoms | 10 | 12
  Grade 3 Headache | 19 | 20
  Grade 3 Myalgia | 10 | 8
  Grade 3 Rash | 0 | 1
  Grade 3 Urticaria | 1 | 2
  Related Arthralgia | 102 | 74
  Related Fatigue | 230 | 181
  Related Fever | 59 | 46
  Related Gastrointestinal symptoms | 134 | 106
  Related Headache | 209 | 187
  Related Myalgia | 132 | 90
  Related Rash | 19 | 11
  Related Urticaria | 24 | 15

17. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.Grade 3 AE = AE that prevented normal activity. Related AE = AE assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 30-day period (Day 0-29) following vaccination
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  Any AEs | 235 | 202
  Grade 3 AEs | 41 | 37
  Related AEs | 70 | 63

18. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs) and Medically Significant Conditions (MSCs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies. MSCs include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: Up to Month 7
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  NOCD(s) | 14 | 13
  MSC(s) | 164 | 148

19. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs) and Medically Significant Conditions (MSCs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies. MSC include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: Up To Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Groups:
- Gardasil Group: Gardasil Group Subjects received 3 doses of Gardasil® (Merck's human papillomavirus [HPV] vaccine) at Months 0, 2 and 6 and a dose of placebo at Month 1. All doses were administered by intramuscular injection in the deltoid muscle of the upper arm.
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  NOCD(s) | 14 | 17
  MSC(s) | 181 | 168

20. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs) and Medically Significant Conditions (MSCs)
Description: as for outcome 19
Time Frame: Up To Month 18
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  NOCD(s) | 20 | 21
  MSC(s) | 210 | 185

21. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs) and Medically Significant Conditions (MSCs)
Description: as for outcome 19
Time Frame: Up To Month 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  NOCD(s) | 20 | 21
  MSC(s) | 221 | 192

22. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs) and Medically Significant Conditions (MSCs)
Description: as for outcome 19
Time Frame: Up To Month 36
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  NOCD(s) | 27 | 29
  MSC(s) | 239 | 205

23. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs) and Medically Significant Conditions (MSCs)
Description: as for outcome 18
Time Frame: Up to Month 48
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  NOCDs | 33 | 33
  MSCs | 251 | 216

24. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs) and Medically Significant Conditions (MSCs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies. MSCs include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
  Note: NOCD and MSC cases were unblinded at the Month 60 analysis.
Time Frame: Up to Month 60
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  Any NOCD(s) | 39 | 43
  Any MSC(s) | 259 | 226

25. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Related SAE = SAE assessed by the investigator as causally related to the study vaccination. Intensity of SAEs was not assessed.
Time Frame: Up to Month 7
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  Any SAE(s) | 6 | 7
  Related SAE(s) | 1 | 1

26. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: as for outcome 25
Time Frame: Up to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  Any SAE(s) | 12 | 20
  Related SAE(s) | 1 | 1

27. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: as for outcome 25
Time Frame: Up to Month 18
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  Any SAE(s) | 14 | 20
  Related SAE(s) | 1 | 1

28. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: as for outcome 25
Time Frame: Up to Month 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  Any SAE(s) | 23 | 22
  Related SAE(s) | 1 | 1

29. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: as for outcome 25
Time Frame: Up to Month 36
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  Any SAE(s) | 30 | 28
  Related SAE(s) | 1 | 1

30. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: as for outcome 25
Time Frame: Up to Month 48
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  Any SAE(s) | 37 | 34
  Related SAE(s) | 1 | 1

31. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Related SAE = SAE assessed by the investigator as causally related to the study vaccination. Intensity of SAE(s) was not assessed.
  Note: SAEs were unblinded at the Month 60 analysis.
Time Frame: Up to Month 60
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Gardasil Group
Number analyzed (Participants) | 553 | 553
Participants
  Any SAE(s) | 44 | 37
  Related SAE(s) | 1 | 1

ADVERSE EVENTS:
Time Frame: SAEs: From Day 0 up to Month 60. Solicited symptoms: During the 7-day (Days 0-6) post-vaccination period.
Description: AEs collected by systematic assessment are reported for subjects with a symptom diary card available. AEs collected non-systematically are reported for the Total Vaccinated Cohort.
Arm/Group | Cervarix Group | Gardasil Group
Serious Adverse Events (participants affected / at risk) | 44/553 | 37/553
Other Adverse Events (participants affected / at risk) | 500/553 | 462/553
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=553) | Gardasil Group (N=553)
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 | 2
Appendicitis (Infections and infestations) | 1 | 2
Menorrhagia (Reproductive system and breast disorders) | 2 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 7 | 4
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 3 | 2
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Major depression (Psychiatric disorders) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Anorexia nervosa (Psychiatric disorders) | 0 | 1
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chest pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Endometritis (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Ileitis (Gastrointestinal disorders) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Spinal shock (Injury, poisoning and procedural complications) | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Uterine enlargement (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=553) | Gardasil Group (N=553)
Pain (General disorders) | 487 | 375
Redness (General disorders) | 232 | 134
Swelling (General disorders) | 191 | 114
Arthralgia (General disorders) | 114 | 81
Fatigue (General disorders) | 262 | 209
Fever (General disorders) | 76 | 58
Gastrointestinal (General disorders) | 172 | 139
Headache (General disorders) | 250 | 220
Myalgia (General disorders) | 145 | 103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.